# **Statistical Analysis Plan (SAP)**

Study No. STP1-C004

A Phase 1b, Double-Blind, Placebo-Controlled, First-in-Human Study to Evaluate Safety, Tolerability and Pharmacokinetics of a Two-Week Oral Treatment with STP1 in a Subgroup of Adult Patients with Autism Spectrum Disorder

Version 1.1

**17 February 2022** 

Prepared for STALICLA SA Campus Biotech Innovation Park Avenue de Secheron 15, 1202 Genève Switzerland

Prepared by STATKING Clinical Services 759 Wessel Drive Fairfield, OH 45014 513-858-2989 www.statkingclinical.com



# **Approval Page**

By entering into this Statistical Analysis Plan (SAP), the parties acknowledge and agree that this SAP shall be incorporated into and subject to the terms of the Master Services Agreement (MSA). Any changes requested by Client to this SAP shall be subject to Section I.C of the MSA requiring a mutually agreed upon "Change Order" prior to any modification of the procedures set forth herein.

I agree to the format and content of this document.

### Approved by:



# Baltazar Gomez-Mancilla, MD, PhD Chief Medical Officer

STALICLA SA Campus Biotech Innovation Park Avenue de Secheron 15, 1202 Genève Switzerland

# Authored by:



Brian Kovacic, PhD Statistician STATKING Clinical Services 759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 301 brian@statkingclinical.com

# Approved by (internal review):

DocuSigned by:

Lori Christman



Signer Name: Lori Christman Signing Reason: I approve this document Signing Time: February 18, 2022 | 10:09 AM EST -D32195A3119A4616B959EFE41655886B

# Lori Christman, PhD Statistician

STATKING Clinical Services 759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 317 lori@statkingclinical.com

# Approved by:

-DocuSigned by:



Signer Name: Mark Tetrick
Signing Reason: I approve this document
Signing Time: February 18, 2022 | 8:58 AM EST
-FF75403BBD93466EABA9DFBDFE59F935

Mark Tetrick, DVM, PhD Clinical Trial Manager STATKING Clinical Services 759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 320

mtetrick@statkingclinical.com

# **Revision History**

# Version 1.0 to 1.1

- SAP updated based on the latest version of the protocol (v6.0)
- Added the cognition crystallized composite results to the in-text description of the NIH Toolbox analysis and to the corresponding table and listing shells in the appendix.
- Updated Section 6.2 to state that the eye tracking data will not be included in the final study database.

# **Table of Contents**

| 1.0 SYNOPSIS OF STUDY DESIGN PROCEDURES | 7 |
|---|---|
| 1.1 Design and Treatment | 7 |
| 1.2 Study Procedures | 8 |
| 1.3 Sample Size | 12 |
| 2.0 DATA ANALYSIS CONSIDERATIONS | 12 |
| 2.1 Types of Analyses | 12 |
| 2.2 Analysis Populations | 13 |
| 2.3 Missing Data Conventions | 13 |
| 2.4 Interim Analyses | 13 |
| 2.5 Study Center Considerations in the Data Analysis | 14 |
| 2.6 Documentation and Other Considerations | 14 |
| 3.0 ANALYSIS OF BASELINE PATIENT CHARACTERISTICS | 14 |
| 4.0 ANALYSIS OF SAFETY | 14 |
| 4.1 Description of Safety Variables | 14 |
| 4.1 Description of Safety Variables | 14 |
| 4.0 ANALYSIS OF SAFETY 4.1 Description of Safety Variables 4.2 Analysis of Safety Variables 5.0 ANALYSIS OF PHARMACOKINETICS 5.1 Description of Pharmacokinetic Variables | 15 |
| 4.1 Description of Safety Variables | 141518 |
| 4.1 Description of Safety Variables | 14<br>15<br>18<br>18 |
| 4.1 Description of Safety Variables | 1415181820 |
| 4.1 Description of Safety Variables | 1415182020 |
| 4.1 Description of Safety Variables | 141518202020 |

| Statistical Analysis Plan | STP1-C004 |
|--------------------------------------------------------|-----------|
| 7.2 Additional Assessments | 23 |
| 7.3 Medical History | 23 |
| 7.4 Concomitant Medication | 23 |
| 8.0 LIST OF ANALYSIS TABLES, FIGURES AND LISTINGS | 24 |
| 9.0 REFERENCES | 29 |
| APPENDIX A – TABLES, FIGURES AND LISTING SPECIFICATION | IS30 |
| APPENDIX B – TABLE SHELLS | 32 |

# 1.0 Synopsis of Study Design Procedures

This study is a randomized, double-blind, placebo-controlled, parallel-group, 2-dose ascending study to assess the safety, tolerability, and pharmacokinetics (PK) of 2-week treatment with STP1 (combined doses of ibudilast and bumetanide) in adult patients with idiopathic Autism Spectrum Disorder Phenotype 1 (ASD-Phen1).

The primary objective of this Phase 1b study is to assess the safety and tolerability of 2-week oral treatment twice a day with STP1 in adult individuals with ASD-Phen1. The secondary objective is to determine the plasma pharmacokinetics of ibudilast and bumetanide when given orally in combination, as STP1, for 2 weeks. Additional exploratory objectives will be assessed as outlined in Section 6.0 of this SAP.

This SAP was written in accordance with the Clinical Study Protocol Version 6, Amendment 5. The SAP will be revised if there are future protocol amendments that impact the content included in this document.

# 1.1 Design and Treatment

The first dose cohort (8 eligible patients) will be randomized and allocated to one of two treatment groups using a 3:1 ratio:

- mg oral twice a day (BID) ibudilast mg oral BID bumetanide (N=6)
- Matching oral placebos BID (N=2)

For each dose cohort, the total duration of the study for each patient will be up to 6 weeks, divided as follows:

- A screening phase of up to 2 weeks (from Day -14 to Day -1)
- A double-blind treatment phase of 2 weeks (from Day 1 to Day 14)
- A follow-up phase of 2 weeks after treatment discontinuation (from Day 15 to Day 28)

Once the first cohort (8 patients) finishes 2 weeks of treatment and 2 weeks of follow-up, a Data Safety Monitoring Board (DSMB) will evaluate the safety data to decide whether the dose of ibudilast can be increased as planned to mg, or the study shall be modified or be stopped.

If the DSMB decision supports the start of the next dose level, up to 8 additional eligible patients will be assigned to one of the following two treatment groups (a minimum of 3 patients should be exposed to the highest dose of STP1):

- Image or al BID ibudilast/ 1 mg or al BID bumetanide (up to N=6)
- Matching oral placebos BID (up to N=2)

Patients that participated in the first dose cohort may be allowed to participate in

the second dose cohort if there is no safety concern and after drug washout. Any patient from Cohort 1 that is re-randomized into Cohort 2 will be counted as a new patient in the analysis. That is, re-enrolled patients will be assigned a new patient ID for Cohort 2, re-randomized, and have a new set of CRFs completed.

Figure 1 below summarizes an overview of the study design.



For STP1 dose 2: N= up to 2 placebo and up to 6 STP1 dose 2, randomization is N= up to 8

# 1.2 Study Procedures

The study includes assessments at screening (Days -14 to -1), treatment period (Days 1 to 14), and the follow-up visits (Days 16-18 (optional) and Day 28).

# Screening Period (Visit 1 - Day -14 to Day -1)

Patients will be screened for study eligibility within 14 days prior to treatment (Days -14 to -1). The following screening procedures will be performed:

- Sign an Informed Consent Form (ICF) before any of the study related procedures are performed
- · Eligibility criteria including all inclusion and exclusion criteria
- Record demographics (including age, gender, height, weight, etc.)
- Record medical history including history of substance use
- · Record previous and concomitant medications and therapies
- Measure vital signs (temperature, heart rate (HR), and respiratory rate)
- Orthostatic blood pressure (BP) and HR
- Perform physical examination

- Perform blood laboratory tests (serology, blood chemistry, hematology, and coagulation)
- Perform urinalysis laboratory test
- Perform 12-lead ECG
- Perform urine pregnancy test for women of childbearing potential
- Perform SARS-CoV-2 Test
- Perform alcohol urine test/substance abuse urine test
- Adverse event (AE) assessment and recording
- Perform study-specific assessments: (Suicidality (Columbia Suicide Severity Rating Scale [C-SSRS] or Columbia Classification Algorithm for Suicide Assessment [C-CASA]), Aberrant Behavior Checklist- Second Edition Community (ABC-C), Social Responsiveness Scale, Second Edition (SRS-2), and Stanford Binet Intelligence Scales, Fifth Edition-Abbreviated Battery IQ (SB5 ABIQ), Ohio Autism Clinical Impression Scale -Severity (OACIS-Severity),
   Test of Attentional Performance for Children (KiTAP), Children Sleep habit Questionnaire (CSHQ), Clinical Global Impressions Severity (CGI-S) Scale
  - C-SSRS, OACIS- Severity, NIH-CTB, KiTAP, CSHQ and CGI-S are collected at Screening for only those patients enrolled under Version 4 or subsequent versions of the protocol

# **Treatment Period (Day 1 to Day 14)**

The following procedures will be performed during the treatment period (visits at Day 1, Day 7 & Day 14):

### Visit 2 - Day 1

- Randomization
- Physical examination
- Vital Signs (pre- and post-dose): including temperature, HR, respiratory rate, and BP
- Orthostatic BP assessment (pre- and post-dose)
- ECG-12 lead (pre- and post-dose)
- Substance abuse test (urine)
- Hearing assessment (collected for only those patients enrolled under Version 4 or subsequent versions of the protocol)
- Administration of the study medication
- Study medication supply
- Blood and urine sampling for PK
- Perform study-specific assessments: Suicidality assessment (C-SSRS or C-CASA), OACIS-Severity, NIH-CTB, KiTAP, CSHQ, and CGI-S

- OACIS-Severity and CGI-S are collected for only those patients enrolled under Version 2 or 3 of the protocol. C-SSRS is collected for only those patients enrolled under Version 4 or subsequent versions of the protocol.
- Eye tracking assessment
- EEG (pre- and post-dose)
- Adverse Events
- Previous and Concomitant treatments

# Visit 3 - Day 7

- Physical examination
- Vital Signs: including temperature, HR, and respiratory rate, and BP
- Orthostatic BP assessment
- ECG-12 lead
- Blood sampling for hematology, blood chemistry, and coagulation
- Urine sampling for urinalysis
- · Administration of the study medication and drug accountability
- Blood sampling for PK
- Suicidality assessment (C-SSRS or C-CASA) (C-SSRS collected for only those patients enrolled under Version 4 or subsequent versions of the protocol)
- Hearing assessment (collected for only those patients enrolled under Version 4 or subsequent versions of the protocol)
- Adverse Event
- Previous and Concomitant treatments

# **Visit 4 - Day 14**

- Physical examination
- Vital Signs: including temperature, HR, respiratory rate, and BP
- Orthostatic BP assessment
- ECG-12 lead
- Blood sampling for hematology, blood chemistry, and coagulation
- Urine sampling for urinalysis
- · Administration of the study medication and drug accountability
- Blood and urine sampling for PK
- Hearing assessment (collected for only those patients enrolled under Version 4 or subsequent versions of the protocol)
- Perform study-specific assessments: Suicidality (C-SSRS and C-CASA), ABC-C, SRS-2, OACIS-S, Ohio Autism Clinical Impression Scale -Improvement (OACIS - C), KiTAP, CSHQ, Clinical Global Impressions - Improvement (CGI-I) Scale, and CGI-S
  - C-SSRS is collected for only those patients enrolled under Version
     4 or subsequent versions of the protocol.

- Eye tracking assessment
- EEG
- Adverse Events
- Previous and Concomitant treatments

# Visit 5- Day 15 and Optional Visit 6/7/8 - Days 16/17/18

Patients enrolled under Version 2 or 3 of the protocol will have blood and urine PK sampling done 30 hours post Day 14 AM dose (i.e., Day 15). Patients enrolled under Version 4 or subsequent versions of the protocol will be given the option to have their follow-up blood PK sampling visit between Day 16 and Day 18.

- Blood and urine sampling for PK (urine sampling collected for only those patients enrolled under Version 2 or 3 of the protocol)
- Suicidality assessment (C-SSRS, C-CASA) (collected for only those patients enrolled under Version 4 or subsequent versions of the protocol)
- AEs
- Previous and concomitant treatments

# Visit 9- Day 28 - End of Study Follow-Up Visit

Patients who complete the Day 15 study visit or discontinue from the study early will be asked to return to the clinic on Day 28 (± 2 days) for the Follow-up visit. After study completion, AEs should be followed according to the study protocol.

The following procedures will be performed:

- Physical examination
- Vital Signs: including temperature, HR, respiratory rate, and BP
- Orthostatic BP assessment
- ECG-12 lead
- Pregnancy Test (urine) in females
- Blood sampling for hematology, blood chemistry, and coagulation
- Urine sampling for urinalysis
- Drug accountability (if not done at Day 14 visit for only those patients enrolled under Version 4 or subsequent versions of the protocol)
- Blood sampling for PK (collected for only those patients enrolled under Version 2 or 3 of the protocol)
- Perform study-specific assessments: Suicidality (C-SSRS, C-CASA), ABC-C, SRS-2, KiTAP, CSHQ, CGI-I, and CGI-S
  - C-SSRS is collected for only those patients enrolled under Version 4 or subsequent versions of the protocol. SRS-2 is collected for only those patients enrolled under Version 2, 3, or 4 of the protocol.
- Hearing assessment (collected for only those patients enrolled under Version 4 or subsequent versions of the protocol)

- Eye tracking assessment
- EEG
- Adverse Events
- Previous and Concomitant treatments

# 1.3 Sample Size

The target number of patients to be enrolled in this study is up to 16 individuals with ASD-Phen1. Assuming a dropout rate of roughly 20%, the maximum sample size of 20 patients will be enrolled in the study in order to ensure that up to 16 patients (up to 8 per dose level) will have evaluable data after 2 weeks of treatment and 2 weeks of follow-up. They will be randomized with a 3:1 ratio to one of the 2 groups (active/placebo) for each dose level.

Up to six patients per dose level on active and up to two on placebo per dose level is considered sufficient for the primary objective.

# 1.3.1 Replacement of Study Patients

If a patient withdraws from the study after randomization but before receiving any treatment, the next patient randomized will be assigned the same randomization number. This will ensure that the treatment allocation within each treatment group is preserved.

If a patient withdraws from the study after receiving any amount of treatment, the next patient randomized will be assigned to the next available randomization number.

# 2.0 Data Analysis Considerations

# 2.1 Types of Analyses

For this Phase 1b study, descriptive statistics will be provided for all variables by treatment group (placebo data will be pooled from the two dose cohorts). For continuous endpoints, summary statistics, i.e., n (number of non-missing observations), mean, standard deviation (SD), median, minimum, and maximum will be provided. For categorical variables, the frequency count and proportion in each category will be summarized.

As mentioned in Section 1.2 of the SAP, some assessment time points will vary according to which protocol amendment was in place at the time a patient was enrolled. Data from all time points will be summarized as appropriate in accordance with the details provided below in Section 3-7.

All data collected will be presented in the by-patient data listings, sorted by patient and by time point, where appropriate.

# 2.2 Analysis Populations

The following analysis populations will be defined for the study:

**Safety Analysis Population:** The safety population will consist of all patients who have received at least one administration of the study treatments, whether prematurely withdrawn from the study or not. For the safety analysis population, data will be analyzed according to the treatment actually taken.

**Pharmacokinetic (PK) Analysis Population:** The PK population will consist of all patients with at least one administration of the study treatments, and with at least one sample collected and analyzed for plasma drug concentration, whether prematurely withdrawn from the study or not.

**Exploratory Analysis Population:** The Exploratory population will consist of all randomized patients who meet the inclusion/exclusion criteria, received full-course of the study drug as per randomization, have completed the main relevant visits and without any major protocol violations which would render the data unreliable.

Analyses of safety will be performed on the Safety population, as will baseline patient characteristics and demographics. Analysis of PK variables will be performed on the PK population. Analyses of PD data will be performed on the Exploratory population. Prior to the final analysis, a blinded review of the protocol violations will be held in order to determine exclusions from the Exploratory population.

# 2.2.1 Subgroup Definitions

Analyses will be presented by treatment (Imag ibudilast/Imag bumetanide, Imag ibudilast/Imag bumetanide, or placebo (placebo data will be pooled from the two dose cohorts)) as indicated below and shown in Appendix B.

# 2.3 Missing Data Conventions

No missing value imputation will be used. That is, all analyses will be based on the observed data (i.e., complete case analysis).

# 2.4 Interim Analyses

An evaluation of the data by an independent DSMB will take place after 8 patients finish 2 weeks of treatment and 2 weeks of follow-up. The primary responsibilities of the DSMB are to:

1. Review and evaluate the accumulated study data for patient safety, study conduct and progress, and

2. Make recommendation to STALICLA concerning the continuation, modification, or termination of the trial.

Refer to the separate Interim Analysis Plan (IAP) for further details on the interim analyses.

# 2.5 Study Center Considerations in the Data Analysis

A study center is defined as a treatment administration site or group of treatment administration sites under the Placebo and supervision of the same Principal Investigator (PI). This study will be conducted as a single study center, and therefore, study center considerations are not applicable. In case additional site(s) is (are) added with patients enrolled, the SAP will be revised if needed.

### 2.6 Documentation and Other Considerations

The data analyses will be conducted using SAS® Software, version 9.4 or later.

# 3.0 Analysis of Baseline Patient Characteristics

Baseline and demographic characteristics will be summarized by treatment for all patients in the Safety population. Placebo data will be pooled from the two dose groups. Continuous variables will be displayed via summary statistics (n, mean, median, SD, minimum, and maximum). Categorical variables will be summarized via frequency counts and proportions.

A detailed listing of demographics data for each patient will also be provided as shown in Appendix B.

# 4.0 Analysis of Safety

# 4.1 Description of Safety Variables

The safety variables for this study are:

- AEs
- Vital Signs and physical examinations
- FCG
- Clinical Laboratory Parameters
- Hearing Assessment

# 4.2 Analysis of Safety Variables

### **Adverse Events**

Prior to analysis, all AEs will be recorded and classified on the basis of the Medical Dictionary for Regulatory Activities (MedDRA®) terminology. The number and proportion of patients with at least one AE will be summarized by system organ class (SOC) and by preferred term (PT) within SOC for each treatment group.

Similar tables will be provided to display the number and proportion of patients with at least one treatment-related AE, at least one treatment-related AE that led to study treatment discontinuation, at least one serious AE (SAE), at least one treatment-related SAE, at least one treatment-related SAE that led to study treatment discontinuation, at least one AE of special interest (AESI), and at least one AESI that led to study treatment discontinuation by SOC and by PT within SOC. For the purposes of this study, a treatment-related AE is any AE with a relationship to study drug of 'Related'.

In addition, tables will be constructed to summarize AEs by relationship to study drug and by severity.

A separate AE summary table will be constructed to display the number of patients with at least one AE, the number of patients with at least one treatment-related AE, the number of patients with at least one treatment-related AE that led to study treatment discontinuation, the maximum severity of AE by patient, the highest relationship of AE to treatment, the number of patients experiencing at least one SAE, the number of patients with at least one treatment-related SAE, the number of patients with at least one treatment-related SAE that led to study treatment discontinuation, the maximum severity of SAE by patient, the highest relationship of SAE to treatment, the number of patients with at least one AESI, the number of patients with at least one AESI that led to study treatment discontinuation, and the number of deaths.

All AEs will be provided in data listings as shown in Appendix B. AEs having an end date prior to signing the informed consent for this study will not be displayed in the AE data listings.

### **Vital Signs**

The vital signs parameters of interest include temperature, respiratory rate, and orthostatic blood pressure and orthostatic heart rate.

Summary statistics (n, mean, median, SD, minimum, and maximum) will be computed on the raw and change from baseline values for standard vital sign measurements (temperature and respiratory rate) by visit and time for each treatment. The Day 1 prior to treatment time point will serve as baseline. If there are multiple vital signs taken at any time point, then the latest set of vital signs

will be used for the analysis.

Additionally, summary statistics will be computed on the raw and change from baseline values for the orthostatic vital sign measurements (BP and HR) by visit and time for each treatment. The Day 1 prior to treatment time point will serve as baseline. Spaghetti plots of the raw values for orthostatic diastolic BP, orthostatic systolic BP and orthostatic HR will be displayed by patient, time point and treatment.

All vital signs will be provided in data listings as shown in Appendix B. Vital signs taken while standing will be included in the data listings but will not be summarized in the tables.

# **Physical Examination**

All physical examination results will be listed as shown in Appendix B.

### **ECG**

The ECG parameters of interest include HR, PQ, QRS, QT, RR, and QTcF along with information on T and U waves.

As the ECGs are performed in triplicate at Day 1 prior to treatment, the average of the three values for each of the ECG parameters will be used as the baseline value. Summary statistics (n, mean, median, SD, minimum, and maximum) will be computed on the raw and change from baseline values for each parameter by visit and time by treatment and overall. The Day 1 prior to treatment time point will serve as baseline. Spaghetti plots of the raw values for HR and QTcF will be displayed by patient, time point and treatment.

The ECG Interpretations for each of the three ECGs on Day 1 prior to treatment will be used to obtain a Combined Overall ECG Interpretation. The Combined Overall ECG Interpretation in relation to clinical significance at Day 1 prior to treatment (i.e., baseline) will be determined as follows:

- If at least one ECG Interpretation= 'Abnormal clinically significant', then the Combined Overall ECG Interpretation = 'Abnormal clinically significant'.
- Else if there are no readings such that ECG Interpretation = 'Abnormal clinically significant' and there is at least one ECG Interpretation = 'Abnormal not clinically significant', then the Combined Overall ECG Interpretation = 'Abnormal not clinically significant'.
- Else if there are no readings such that ECG Interpretation = 'Abnormal clinically significant' or "Abnormal not clinically significant' and there is at least one ECG Interpretation = 'Normal', then the Combined Overall ECG Interpretation = 'Normal'.
- Else if all readings have a missing result for ECG Interpretation then the Combined Overall ECG Interpretation is missing.

Additionally, results from the ECG findings will be determined for T wave, U wave, and ECG Interpretation regardless of clinical significance. The Combined Overall T wave, U wave, and ECG Interpretation at Day 1 prior to treatment (i.e. baseline) will be determined by parameter as follows:

- If at least one ECG finding = 'Abnormal', then the Combined Overall finding = 'Abnormal'.
- Else if there are no readings such that ECG finding = 'Abnormal' and there is at least one ECG finding = 'Normal', then the Combined Overall finding = 'Normal'.
- Else if all readings have a missing result for ECG finding then the Combined Overall finding is missing.

Shift tables will be constructed to show the changes in ECG findings in relation to clinical significance (e.g., normal, abnormal clinically significant (CS), abnormal not clinically significant (NCS)) and findings (e.g., normal, abnormal) by parameter from baseline to each visit by treatment and overall.

All ECG data will be provided in data listings as shown in Appendix B.

# **Laboratory Results**

The laboratory tests of interest include blood chemistry, serology, hematology, coagulation, and urinalysis results.

Summary statistics (n, mean, median, SD, minimum, and maximum) will be computed on the raw and change from baseline values for each quantitative laboratory parameter by visit for each treatment group and overall. The screening time point will serve as baseline.

Spaghetti plots of the raw values for sodium, chloride, calcium, magnesium, phosphate, potassium, and platelet count will be displayed by patient, time point and treatment.

For those urinalysis parameters that are qualitative in nature, the number and proportion of patients with each result for each parameter will be summarized by visit and treatment.

Shift tables will be constructed to show the changes in laboratory results in relation to clinical significance (e.g., normal, abnormal clinically significant (CS), abnormal not clinically significant (NCS)) from baseline to each visit. This analysis will be repeated for blood chemistry results for electrolytes (sodium, chloride, calcium, magnesium, phosphate, potassium).

A shift table for blood chemistry results for electrolytes will be constructed to show the changes in laboratory results in relation to range of normal results (e.g., normal, high, low) from baseline to each visit.

The count and proportion of patients with blood chemistry results for electrolytes outside of the normal range (low, high) for each visit will be summarized by treatment and overall.

All laboratory results data will be provided in data listings as shown in Appendix B.

# **Hearing Assessment**

The patient responses to the hearing assessment for each visit will be listed as shown in Appendix B.

# 5.0 Analysis of Pharmacokinetics

# 5.1 Description of Pharmacokinetic Variables

PK sampling will be collected from all patients for measurement of plasma and urine concentrations of ibudilast and bumetanide.

Blood samples will be drawn on Days 1, 7, 14/15 and, optionally, between Days 16 to 18, and urine samples will be collected on Days 1 and 14 to determine concentrations of ibudilast and bumetanide. Non-compartmental analysis (NCA) will be utilized to analyze data from the sampling schema. See Table 1 for the PK sample schedule.

| PK Schedule <sup>c</sup> | | |
|---|---|---|
| Time | Plasma <sup>a</sup> | Urine <sup>b</sup> |
| Day 1 | 0.25, 0.5, 1, 2, 4, and 6h post-AM dose | 0 to 6h post-AM dose |
| Day 7 | Pre-AM dose | |
| Day 14 (only AM | Pre-AM dose and 0.25, 0.5, 1, 2, 4, 6, 8, 10, 12 | 0 to 4h, 4 to 8h, and |
| dose) and 15 | and 24h post-AM dose | 8-12h post-AM dose |
| Between Days 16 | 48, 72, and 96 h post-AM dose of Day 14 | |
| to 18 <sup>d</sup> | | |
| a Poth inuditact and humotonide will be analyzed from the same blood draw for each | | |

**Table 1. PK Sampling Schedule** 

The following PK plasma parameters will be estimated for each patient(as far as possible):

<sup>&</sup>lt;sup>a</sup> Both ibudilast and bumetanide will be analyzed from the same blood draw for each specified sampling time point.

<sup>&</sup>lt;sup>b</sup> Urine creatinine from the urine collection will be paired with a serum creatinine measurement to evaluate completeness of collection.

<sup>&</sup>lt;sup>c</sup> All of these timepoints have a 5-minute window.

<sup>&</sup>lt;sup>d</sup> Optional

| PK Parameter | Definition |
|---|---|
| Cmax, Day 1 | Maximum plasma concentration on Day 1 |
| C <sub>max,ss</sub> | Maximum plasma concentration at steady state |
| CLast | Last measured plasma concentration following |
| | the last administration |
| Ctrough | Minimum observed plasma concentration prior |
| | to drug administration |
| T <sub>max</sub> | Time of maximum observed plasma |
| | concentration; if it occurs at more than one time |
| | point, T <sub>max</sub> is defined as the first time point with |
| | this value |
| t <sub>1/2</sub> | Terminal elimination half-life, calculated as |
| | In(2)/λz |
| AUC <sub>0-last</sub> | Cumulative area under the plasma concentration |
| | time curve calculated from 0 to the last |
| | measured plasma concentration following the last administration using the linear trapezoidal |
| | method |
| AUC <sub>0-tau</sub> (6h), Day 1 | Area under the plasma concentration time |
| 7 to So-tau (OII), Day 1 | curve to the end of the dosing period following |
| | the first administration |
| AUC <sub>0-tau</sub> (6h), SS | Area under the plasma concentration time |
| ` ' | curve to the end of the dosing period (6h) |
| | following the last administration |
| AUC <sub>0-12h</sub> , ss | Area under the plasma concentration time |
| | curve to 12 hours post dose following the last |
| | administration |
| AUC <sub>0-∞</sub> | Area under the plasma concentration time |
| | curve extrapolated to infinity, calculated as |
| | AUC <sub>0-last</sub> + C <sub>Last</sub> /λz |
| Vz/F | Apparent volume of distribution |
| CI/F | Apparent total body clearance |
| Accumulation Ratio | Ratio of accumulation of a drug, calculated by |
| | the following equation: |
| | ARAUC = AUC0-tau (6h), ss / AUC0-tau (6h), Day 1 |
| | and ARcmax = Cmax,ss / Cmax, Day 1 |

As the PK time schedules were different prior to the implementation of Version 4.0 (Amendment 3) of the clinical study protocol, the PK schedule of the first 4 patients is as follows:

# Day 1

- Blood sampling at pre-AM dose and 0.25, 0.5, 1, 2, 4, 6 h post-AM dose
- Urine sampling at 0 to 6 h post-AM dose

# Day 7

Blood sampling at pre-AM dose

# Day 14

- Blood sampling at pre-AM dose and 0.25, 0.5, 1, 2, 4, 6, 8, 10, 24 and 30 h post-AM dose
- Urine sampling 0 to 6 h and 24 to 30 h post-AM dose

# 5.2 Analysis of Pharmacokinetic Variables

Plasma and urine sample concentrations of ibudilast and bumetanide will be summarized by treatment, visit and time point using descriptive statistics.

Individual plasma concentrations of ibudilast and bumetanide will be depicted for each patient by treatment group using linear scale. Individual and mean plasma concentration- time profiles will be plotted in linear and semi-logarithmic scales.

PK parameter values will be summarized by treatment group using descriptive statistics (n, mean, SD, CV%, geometric mean, and 90% confidence interval). Plasma PK parameters such as AUC<sub>0-tau</sub>, AUC<sub>last</sub>, C<sub>max</sub>, T<sub>max</sub>, C<sub>trough</sub>, apparent oral clearance, the elimination half-life, apparent volume of distribution and accumulation ratios will be calculated following single dose administration (as far as possible) and at steady state for both parent drugs.

Urine parameters include the following:

- Excretion rate by timepoint:
  - o Day 1, 0-6h
  - o Day 14, 0-4h
  - o Day 14, 4-8h
  - o Day 14, 8-12h
- Cumulative excretion, based on Day 14 sampling over 0-12h
- Renal clearance, based on Day 14 sampling over 0-12h

# 6.0 Exploratory Analyses

# 6.1 Description of Exploratory Variables

Exploratory variables for this study include:

- and KiTAP subtask score
- OACIS-C
- ABC-C subscale scores
- SRS-2 subscale scores
- CSHQ total score
- Lactate and Pyruvate Blood Levels
- Change from baseline in CGI-S, as reflected by CGI-I
- Eye tracking
- EEG

# 6.2 Analysis of Exploratory Variables

# and KiTAP

Summary statistics (n, mean, median, SD, minimum, and maximum) will be computed on the raw and change from baseline values for each subtask variable by visit, treatment and overall. The Day 1 time point will serve as baseline.

### **OACIS-C**

Summary statistics (n, mean, median, SD, minimum, and maximum) will be computed on the raw score for each question will be summarized by treatment and overall. Frequency counts and proportions will also be summarized for each response in the assessment by treatment and for each group of responses (very much improved or much improved; minimally improved, no change or minimally worse; and much worse or very much worse).

### ABC-C

Summary statistics (n, mean, median, SD, minimum, and maximum) will be computed on the raw and change from baseline scores for each subscale by visit, treatment and overall. The Screening time point will serve as baseline.

### SRS-2

Summary statistics (n, mean, median, SD, minimum, and maximum) will be computed on the raw and change from baseline scores for each subscale by visit, treatment and overall. The Screening time point will serve as baseline.

### **CSHQ**

The number and proportions will be summarized for each value in the assessment by visit, question, treatment and overall. The Day 1 time point will serve as baseline.

# **Lactate and Pyruvate Blood Levels**

Summary statistics (n, mean, median, SD, minimum, and maximum) will be computed on the raw and change from baseline values of lactate, pyruvate and lactate-pyruvate ratio (L:P ratio) by treatment and overall. The Screening time point will serve as baseline.

Spaghetti plots of the raw values for L:P ratio will be displayed by patient, time point and treatment.

# CGI-S and CGI-I

Frequency counts and proportions for each response to the CGI-S and CGI-I assessments will be summarized by treatment and visit. Patients enrolled under

protocol Version 3 or earlier will be summarized at the following visits: Days 1, 14 and 28. Patients enrolled under Version 4 or later will be summarized at the following visits: Screening, Days 14 & 28. Data will be combined for overlapping visits.

# **Eye Tracking and EEG**

Eye tracking will not be included in the final study database. However, EEG data will be included in the final study database.

Both the eye tracking and EEG data will not be incorporated into the analysis datasets nor the tables, listings, and figures covered in this SAP. Analysis plans for the eye tracking and EEG variables will be presented in a separate document. The variables to be analyzed to assess changes from Day 1 to Day 14 are as follows:



Eye Tracking variables:

- 1. Time spent mouth and eyes
  - a. Region
  - b. Total time

# 7.0 Other Relevant Data Analyses/Summaries

# 7.1 Patient Disposition

A table will be constructed with the number of screen failures and enrolled patients. For those patients who are screen failures, the number and proportion for each reason for screen failure will be summarized. Of those enrolled, frequency counts and proportion of the number of patients withdrawing from the study before study completion and the number completing the study will be displayed. For those patients that withdraw before completion of the study or discontinue treatment of STP1, the number and proportion for each reason for withdrawal will be tabulated. The table will include summary counts and proportions by treatment and overall. A data listing of all patient completion and withdrawal data will also be constructed.

# 7.2 Additional Assessments

Suicidality (C-SSRS, C-CASA) assessments will be performed at Screening, throughout the treatment period and at the follow-up visits, as specified in the protocol. The SB5 ABIQ assessment will be completed at Screening only. These assessments will be listed for all patients in the Safety population as shown in Appendix B.

# 7.3 Medical History

Prior to analysis, all medical history terms will be coded using the MedDRA coding dictionary. The number and proportion of patients with at least one medical history term will be summarized by system organ class (SOC) and by preferred term (PT) within SOC for each treatment group.

A complete medical history of past and present illnesses and surgeries will be listed as shown in Appendix B.

# 7.4 Concomitant Medication

All concomitant medications will be coded with the WHO Drug Dictionary. A table will be constructed with number and proportion of patients by ATC level 4 and preferred term.

All concomitant medications will be listed as shown in Appendix B.

# 8.0 List of Analysis Tables, Figures and Listings

| Table<br>No. | Table Title | Included<br>in Final<br>Tables | Shown in<br>Appendix<br>B |
|---|---|---|---|
| | 1,50,000 | 10.0.00 | |
| 1 | Patient Disposition | | Х |
| 2 | Demographics and Baseline Data Summary Statistics–<br>Continuous Variables (Safety Population) | Х | Х |
| 3 | Demographics and Baseline Data Summary Statistics–<br>Categorical Variables (Safety Population) | Х | Х |
| 4 | Summary of Adverse Events (Safety Population) | Х | Х |
| 5 | Number and Proportion of Patients with Adverse Events (Safety Population) | Х | Х |
| 6 | Number and Proportion of Patients with Treatment-<br>Related Adverse Events (Safety Population) | Х | Х |
| 7 | Number and Proportion of Patients with Treatment-<br>Related Adverse Events that Led to Study Drug<br>Discontinuation (Safety Population) | х | х |
| 8 | Number and Proportion of Patients with Serious Adverse Events (Safety Population) | Х | Х |
| 9 | Number and Proportion of Patients with Treatment-<br>Related Serious Adverse Events (Safety Population) | х | Х |
| 10 | Number and Proportion of Patients with Treatment-<br>Related Serious Adverse Events that Led to Study Drug<br>Discontinuation (Safety Population) | Х | Х |
| 11 | Number and Proportion of Patients with Adverse Events of Special Interest (Safety Population) | Х | Х |
| 12 | Number and Proportion of Patients with Adverse Events of Special Interest that Led to Study Drug Discontinuation (Safety Population) | Х | Х |
| 13 | Number and Proportion of Patients with Adverse Events by Relationship to Study Drug (Safety Population) | Х | Х |
| 14 | Number and Proportion of Patients with Adverse Events by Severity (Safety Population) | Х | Х |
| 15 | Vital Sign Parameter Summary Statistics (Safety Population) | Х | Х |
| 16 | Orthostatic Vital Sign Parameter Summary Statistics (Safety Population) | X | Х |
| 17 | ECG Parameter Summary Statistics (Safety Population) | X | X |
| 18 | ECG Results Shift Table by Visit and Clinical Significance (Safety Population) | X | Х |
| 19 | ECG Results Shift Table by Visit (Safety Population) | Х | Х |
| 20 | Blood Chemistry Parameter Summary Statistics (Safety Population) | Х | Х |
| 21 | Hematology Parameter Summary Statistics (Safety Population) | Х | |
| 22 | Coagulation Parameter Summary Statistics (Safety Population) | х | |
| 23 | Quantitative Urinalysis Parameter Summary Statistics (Safety Population) | Х | |
| 24 | Summary of Qualitative Urinalysis Results by Parameter (Safety Population) | Х | Х |

| Table<br>No. | Table Title | Included<br>in Final<br>Tables | Shown in<br>Appendix<br>B |
|---|---|---|---|
| 25 | Blood Chemistry Results Shift Table by Visit and Clinical | Х | Х |
| | Significance (Safety Population) | ^ | ^ |
| 26 | Hematology Results Shift Table by Visit and Clinical | Х | |
| | Significance (Safety Population) | ^ | |
| 27 | Coagulation Results Shift Table by Visit and Clinical | X | |
| | Significance (Safety Population) | | |
| 28 | Quantitative Urinalysis Results Shift Table by Visit and Clinical Significance (Safety Population) | X | |
| 29 | Blood Chemistry Results for Electrolytes Shift Table by | | |
| | Visit and Clinical Significance (Safety Population) | X | |
| 30 | Blood Chemistry Results for Electrolytes Shift Table by | | |
| | Visit and Range of Normal Results (Safety Population) | X | X |
| 31 | Number and Proportion of Patients with Blood | | |
| | Chemistry Results for Electrolytes Outside of Normal | X | X |
| | Range (Safety Population) | | |
| 32 | Summary Statistics of Ibudilast and Bumetanide Plasma | | |
| | Concentration Levels by Treatment, Visit and Time (PK | X | X |
| | Population) | | |
| 33 | Summary Statistics of Ibudilast and Bumetanide Urine | | |
| | Concentration Levels by Treatment, Visit and Time (PK | X | X |
| | Population) | | |
| 34 | Summary Statistics of Estimated PK Plasma | X | Х |
| | Parameters for Ibudilast by Treatment (PK Population) | ^ | ^ |
| 35 | Summary Statistics of Estimated PK Plasma | | |
| | Parameters for Bumetanide by Treatment (PK | X | X |
| | Population) | | |
| 36 | Summary Statistics of Estimated PK Urine Parameters | X | × |
| | for Ibudilast by Treatment (PK Population) | | , |
| 37 | Summary Statistics of Estimated PK Urine Parameters | X | |
| | for Bumetanide by Treatment (PK Population) | | |
| 38 | | X | X |
| 39 | KiTAP Summary Statistics (Exploratory Population) | X | |
| 40 | OACIS-C Summary Statistics (Exploratory Population) | X | X |
| 41 | Summary of Responses for OACIS-C Assessment by | X | × |
| 40 | Question (Exploratory Population) | , , | |
| 42 | Summary of Responses for OACIS-S Assessment by | X | X |
| 40 | Question (Exploratory Population) | | |
| 43 | ABC-C Summary Statistics (Exploratory Population) | X | X |
| 44 | SRS-2 Summary Statistics (Exploratory Population) | | |
| 45 | Summary of Responses for CSHQ Assessment by | X | × |
| 40 | Question (Exploratory Population) | | |
| 46 | Lactate and Pyruvate Blood Level Summary Statistics | X | × |
| 47 | (Exploratory Population) | | , , |
| 47 | Summary of Responses for CGI-S Assessment by Visit | X | × |
| | (Exploratory Population) Summary of Responses for CGI-I Assessment by Visit | | |
| 40 | I Summary of Responses for CGI-L Assessment by Visit | 1 | I |
| 48 | | X | X |
| 48 | (Exploratory Population) Number and Proportion of Patients with Medical History | X | X |

| Table<br>No. | Table Title | Included<br>in Final<br>Tables | Shown in<br>Appendix<br>B |
|---|---|---|---|
| 50 | Number and Proportion of Patients Taking Concomitant Medications by ATC Level 4 and Preferred Term (Safety Population) | x | X |

| No. | Listing Title | Listings | Shown in Appendix B |
|---|---|---|---|
| DL1 | Patient Disposition Data Listing | Х | X |
| DL2 | Demographics Data Listing | Х | X |
| DL3 | Adverse Events Data Listing | Х | X |
| DL4 | Vital Signs Data Listing | X | Х |
| DL5 | Baseline ECG Data Listing | X | Х |
| DL6 | ECG Data Listing | Х | X |
| DL7 | Blood Chemistry Laboratory Results Data Listing | Х | X |
| DL8 | Serology Laboratory Results Data Listing | Х | Х |
| DL9 | Hematology Laboratory Results Data Listing | Х | X |
| DL10 | Coagulation Laboratory Results Data Listing | Х | |
| DL11 | Urinalysis Laboratory Results Data Listing | Х | |
| DL12 | Hearing Assessment Data Listing | Х | Х |
| DL13 | Pharmacokinetic Blood Sample Data Listing | Х | Х |
| DL14 | Pharmacokinetic Urine Sample Data Listing | Х | Х |
| DL15 | Plasma Concentrations Data Listing | Х | Х |
| DL16 | Urine Concentrations Data Listing | Х | Х |
| DL17 | Plasma Pharmacokinetics Parameters Data Listing | Х | X |
| DL18 | Urine Pharmacokinetics Parameters Data Listing | Х | X |
| DL19 | C-SSRS Data Listing | X | X |
| DL20 | C-CASA Data Listing | Х | Х |
| DL21 | OACIS-S Data Listing | Х | X |
| DL22 | OACIS-C Data Listing | X | X |
| DL23 | SRS-2 Data Listing | Х | X |
| DL24 | SB5 ABIQ Data Listing | Х | X |
| DL25 | | X | X |
| DL26 | KiTAP Data Listing | X | + |
| DL27 | ABC-C Data Listing | X | X |
| DL28 | CSHQ Data Listing | X | X |
| DL29 | Lactate-Pyruvate Data Listing | X | X |
| DL30 | CGI-S/CGI-I Data Listing | X | X |
| DL31 | Medical History Data Listing | Х | X |
| DL32 | Concomitant Medications Data Listing | X | X |
| DL33 | Physical Exam Data Listing | X | X |
| DL34 | Study Drug Administration Data Listing | X | X |
| DL35 | Drug Accountability Data Listing | X | X |
| DL36 | Urine Pregnancy Test Data Listing | X | X |
| DL37 | Protocol Deviations Data Listing | X | X |
| DL38 | Patients Excluded from Safety Population Data Listing | X | X |
| DL39 | Patients Excluded from PK Population Data Listing | Х | 1 |

| Listing<br>No. | Listing Title | Included<br>in Final<br>Listings | Shown in<br>Appendix B |
|---|---|---|---|
| DL40 | Patients Excluded from Exploratory Population Data Listing | X | |

| Figure<br>No. | Figure Title | Included<br>in Final<br>Listings | Shown in<br>Appendix B |
|---|---|---|---|
| | | | - 4- p |
| FIG1 | Orthostatic Vital Signs - Spaghetti Plot of Systolic<br>Blood Pressure by Patient, Time and Treatment<br>(Safety Population) | Х | Х |
| FIG2 | Orthostatic Vital Signs - Spaghetti Plot of Diastolic<br>Blood Pressure by Patient, Time and Treatment<br>(Safety Population) | X | |
| FIG3 | Orthostatic Vital Signs - Spaghetti Plot of Heart<br>Rate by Patient, Time and Treatment (Safety<br>Population) | X | |
| FIG4 | ECG Parameters - Spaghetti Plot of Heart Rate by Patient, Time and Treatment (Safety Population) | Х | |
| FIG5 | ECG Parameters - Spaghetti Plot of QTcF by Patient, Time and Treatment (Safety Population) | Х | |
| FIG6 | Blood Chemistry - Spaghetti Plot of Sodium by Patient, Time and Treatment (Safety Population) | Х | Х |
| FIG7 | Blood Chemistry - Spaghetti Plot of Chloride by Patient, Time and Treatment (Safety Population) | Х | |
| FIG8 | Blood Chemistry - Spaghetti Plot of Calcium by Patient, Time and Treatment (Safety Population) | Х | |
| FIG9 | Blood Chemistry - Spaghetti Plot of Magnesium by Patient, Time and Treatment (Safety Population) | Х | |
| FIG10 | Blood Chemistry - Spaghetti Plot of Phosphate by Patient, Time and Treatment (Safety Population) | Х | |
| FIG11 | Blood Chemistry - Spaghetti Plot of Potassium by Patient, Time and Treatment (Safety Population) | Х | |
| FIG12 | Hematology - Spaghetti Plot of Platelet Count by Patient, Time and Treatment (Safety Population) | Х | |
| FIG13 | Biomarker - Spaghetti Plot of L:P Ratio by Patient,<br>Time and Treatment (Safety Population) | Х | |
| FIG14 | Patient Plasma Concentration Levels of Ibudilast for Treatment Group = mg Ibudilast – Linear Scale – Days 1-28 (PK Population) | Х | Х |
| FIG15 | Patient Plasma Concentration Levels of Ibudilast for Treatment Group = mg Ibudilast Linear Scale – Days 1-28 (PK Population) | Х | |
| FIG16 | Patient Plasma Concentration Levels of Ibudilast for Treatment Group = mg Ibudilast – Semi-Logarithmic Scale – Days 1-28 (PK Population) Patient Plasma | Х | |
| FIG17 | Concentration Levels of Ibudilast for Treatment Group = mg Ibudilast – Semi-Logarithmic Scale – Days 1-28 (PK Population) | Х | |

| Figure | | Included in Final | Shown in |
|---|---|---|---|
| No. | Figure Title | Listings | Appendix B |
| FIG18 | Patient Plasma Concentration Levels of | X | |
| | Bumetanide for Treatment Group = mg Ibudilast- | | |
| F10.10 | Linear Scale – Days 1-28 (PK Population) | | |
| FIG19 | Patient Plasma Concentration Levels of | X | |
| | Bumetanide for Treatment Group = mg Ibudilast- | | |
| FIG20 | Linear Scale – Days 1-28 (PK Population) Patient Plasma Concentration Levels of | X | |
| FIG20 | Bumetanide for Treatment Group = Img Ibudilast | ^ | |
| | Semi-Logarithmic Scale – Days 1-28 (PK | | |
| | Population) | | |
| FIG21 | Patient Plasma Concentration Levels of | X | |
| 11021 | Bumetanide for Treatment Group = mg Ibudilast- | | |
| | Semi-Logarithmic Scale – Days 1-28(PK | | |
| | Population) | | |
| FIG22 | Mean Plasma Concentration Levels of Ibudilast for | X | X |
| | Treatment Group = mg Ibudilast – Linear Scale – | | |
| | Days 1-28 (PK Population) | | |
| FIG23 | Mean Plasma Concentration Levels of Ibudilast for | Х | |
| | Treatment Group = mg Ibudilast – Linear Scale – | | |
| | Days 1-28 (PK Population) | | |
| FIG24 | Mean Plasma Concentration Levels of Ibudilast for | X | |
| | Treatment Group = mg Ibudilast – Semi- | | |
| | Logarithmic Scale – Days 1-28 (PK Population) | | |
| FIG25 | Mean Plasma Concentration Levels of Ibudilast for | X | |
| | Treatment Group = mg Ibudilast – Semi- | | |
| | Logarithmic Scale – Days 1-28 (PK Population) | | |
| FIG26 | Mean Plasma Concentration Levels of Bumetanide | X | |
| | for Treatment Group = mg Ibudilast – Linear Scale | | |
| FI007 | – Days 1-28 (PK Population) | | |
| FIG27 | Mean Plasma Concentration Levels of Bumetanide | Х | |
| | for Treatment Group = mg Ibudilast – Linear | | |
| FIG28 | Scale – Days 1-28 (PK Population) Mean Plasma Concentration Levels of Bumetanide | | |
| FIGZŐ | for Treatment Group = mg Ibudilast – Semi- | X | |
| | Logarithmic Scale – Days 1-28 (PK Population) | | |
| FIG29 | Mean Plasma Concentration Levels of Bumetanide | X | |
| 1 1028 | for Treatment Group = mg Ibudilast – Semi- | ^ | |
| | Logarithmic Scale – Days 1-28 (PK Population) | | |
| | Logarianino Codio Dayo 1-20 (1 K 1 opulation) | 1 | |

# 9.0 References

Not applicable.

# **Appendix A – Tables, Figures and Listing Specifications**

### Orientation

Tables, figures, and listings will be displayed in landscape.

# **Margins**

Margins will be 1 inch on all sides. Table, figure, and listing boundaries will not extend into the margins.

### **Font**

Courier New, 8 point.

### **Headers**

The table number will be on the second line of the title area. The title area will contain the Sponsor name, the study number, and the name of the table. The title area will contain the page number (Page x of y) on the far right, one line above the name of the table.

### **Footers**

- The first line will be a solid line.
- Next will be any footnotes regarding information displayed in the table.
- Below these footnotes will be displayed "STATKING Clinical Services (month day, year)" on the far left.
- The last line will display the name of the SAS program that generated the table and (if applicable) the source data reference.

### **Table Disclaimer**

The format of the mock tables shown in the appendix of this Statistical Analysis Plan (SAP) will be the format of the deliverable tables to the extent that Word document constructed tables can match production tables produced by SAS. This formatting includes the content and format of the header and footer areas of the tables. The Sponsor agrees to the format of the tables as shown in the appendix.

Further programming charges will be applicable for changes in the format of tables (including title statements, notes, data dependent footnotes, etc.) made after the approval of the SAP.

# **Missing Values**

All missing values will be displayed on the output tables/listings as blanks.

# **Computation Values for Study Dates**

The date format to be used is dd-mmm-yyyy. Missing parts of dates are not shown (e.g., for a missing day value, the value displayed is in mmm-yyyy format).

# Appendix B – Table Shells

Tab

| CLA | ole |
|-----------|-------------|
| SA | |
| 1 | Pa |
| Study | Patient |
| No. | Disp |
| STP1-C004 | Disposition |

Page x of y

| Reason for Discontinuation from STP1 Pregnancy Patient Non-compliance Patient Unblinding xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Reason for Patient Discontinuation Adverse Event Investigator Decision Consent Withdrawn Patient Non-compliance Death Other | Completed Discontinued | Enrolled | Reason for Screen Failure xxxxxxxxxxxxxxxxxxx xxxxxxxxxxxxxx | Screen Failures |
|---|---|---|---|---|---|
| * * * * * | * * * * * * * | × × | | | STP:<br>ibu |
| (xxx)<br>(xxx)<br>(xxx)<br>(xxx) | ( | (xxx) | × | | STP1-XX ibudilast (N=xxx) a |
| × | × | × × | | | STP<br>ibu |
| ( | ( | (xxx) | ×× | | ibudilast (N=xxx) a |
| | $\begin{smallmatrix} \times & \times & \times & \times & \times \\ \times & \times & \times & \times & \times \\ \times & \times &$ | × × | | | P1 |
| | ( | (xxx) | × | | Placebo<br>(N=xxx) ª |
| × | × | × × | | | Ove |
| ( | ( | xxx (xxx) | × | * * * | Overall (N=xxx) |

The denominator for all proportions is the number of enrolled patients in the corresponding treatment group and overall. STATKING Clinical Services (month day, year)
Source Program: xxxxxxx.sas

Table 2. Demographics and Baseline Data Summary Statistics - Continuous Variables STALICIA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| SB5-ABIQ | | ВМІ | Weight (kg) | Height (cm) | Age (years) | Variable |
|---|---|---|---|---|---|---|
| STP1 mg ibudilast STP1 mg ibudilast Placebo Overall | STP1-Xmg ibudilast STP1-Xmg ibudilast Placebo Overall | STP1 mg ibudilast STP1 mg ibudilast STP1 mg ibudilast Placebo Overall | STP1- mg ibudilast STP1- mg ibudilast Placebo | STP1—— ng ibudilast<br>STP1—— ng ibudilast<br>Placebo<br>Overall | STP1-\(\text{mg ibudilast}\) STP1-\(\text{mg ibudilast}\) Placebo Overall | Treatment Group |
| × | × | × | | × | × × × ×<br>× × × × | n |
| × | × | * | | × | × × × ×<br>× × × × | Mean |
| × | × | × | : | × | × × × ×<br>× × × × | Std Dev |
| × | * * * * * | × | | × | × × × ×<br>× × × × | Median |
| × | × | × | | × | × | Min |
| × | × | × | | × | × × × ×<br>× × × × | Max |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Table 3. Demographics and Baseline Data Summary Statistics - Categorical Variables STALICIA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| Ethnicity | | | | | Race | | Sex | Demographics<br>Variable |
|---|---|---|---|---|---|---|---|---|
| Hispanic<br>Not Hispanic | Other | Hawaiian<br>White | Black | Asian | American Indian | Female | Male | Category |
| × ×<br>× × | XXX | × ×<br>× × | ××× | ××× | ××× | ××× | ××× | ibu<br>(N |
| (xxx)<br>(xxx) | (XXX) | ( | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | STP1mg<br>ibudilast<br>(N=xxx) <sup>a</sup> |
| × × × × | ××× | × ×<br>× × | ××× | ××× | ××× | ××× | ××× | STP1<br>ibu<br>(N= |
| (xxx)<br>(xxx) | (xxx) | ( | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | ibudilast (N=xxx) <sup>a</sup> |
| × × × × | XXX | × ×<br>× × | ××× | ××× | ××× | ××× | ××× | P1a<br>(N= |
| (xxx)<br>(xxx) | (xxx) | ( | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | Placebo<br>(N=xxx) <sup>a</sup> |
| × ×<br>× × | ××× | × ×<br>× × | ××× | ××× | ××× | ××× | ××× | Ove |
| ( | (xxx) | ( | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | Overall (N=xxx) a |

The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall. STATKING Clinical Services (month day, year)
Source Program: xxxxxxx.sas


Table 4. Summary of Adverse Events STALICLA SA - Study No. STP1-C004 Safety Population (N=xxxx)

Page x of y

| STP | $STP1-Mmg$ ibudilast $(N=xxx)^a$ | $STP1-\underset{(N=xxx)^a}{\underbrace{\hspace{1.5cm}}}$ ng ibudilast | Placebo<br>(N=xxx) <sup>a</sup> | Overall (N=xxx) a |
|---|---|---|---|---|
| Patients with at Least One Adverse Event (AE) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Patients with at Least One Treatment-Related AE | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Patients with at Least One Treatment-Related AE that<br>Led to Study Treatment Discontinuation | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Maximum AE Severity Grade | | | | |
| Mild | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Moderate | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Severe | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Highest Relationship of AE to Study Drug | | | | |
| Not Related | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Related | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Patients with at Least One Serious AE (SAE) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Patients with at Least One Treatment-Related SAE | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Patients with at Least One Treatment-Related SAE that Led to Study Treatment Discontinuation | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| [Table continues on next page.] | | | | עק |

The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall. STATKING Clinical Services (month day, year) Source Program: xxxxxxxx.sas

STATKING Clinical Services Version 1.1
Table 4. Summary of Adverse Events STALICLA SA - Study No. STP1-C004 Safety Population (N=xxxx)

Page x of y

| Patients with at Least One AE of Special Interest xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) (AESI) Patients with at Least One AESI that Led to Study xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) Treatment Discontinuation xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) | Maximum SAE Severity Grade Mild Moderate Severe Highest Relationship of SAE to Study Drug Not Related Related | XTP1- mg ibudilast (N=xxx)* xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) | STP1-Mag ibudilast STP1-Mag ibudilast (N=xxx)** xxx (xxx) | Placebo (N=xxx) <sup>a</sup> xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) | Overall (N=xxx) <sup>a</sup> xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) |
|---|---|---|---|---|---|
| XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) | Moderate<br>Severe | xxx (xxx) xxx | xxx (xxx) | xxx (xxx) | xxx (xxx)<br>xxx (xxx) |
| XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) | Highest Relationship of SAE to Study Drug | | | | |
| XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) XXX (XXX) | Not Related | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) | Related | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| AESI that Led to Study xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) | Patients with at Least One AE of Special Interest (AESI) $$ | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| xxx (xxx) xxx (xxx) xxx (xxx) | | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| | Deaths | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |

The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall. STATKING Clinical Services (month day, year)
Source Program: xxxxxxx.sas


Table 5. Number and Proportion of Patients with Adverse Events STALICLA SA - Study No. STP1-C004
Safety Population (N=xxx)

Page x of y

| Preferred Term 2 | Preferred Term 1 | System Organ Class 2 | Preferred Term 2 | Preferred Term 1 | System Organ Class 1 | Patients with at Least One AE | Total Number of Adverse Events (AEs) | Adverse Event Categoryª: |
|---|---|---|---|---|---|---|---|---|
| xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | ××× | STP1-Xmg<br>ibudilast<br>(N=xxx) <sup>b</sup> |
| xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | ××× | STP1-\_mg ibudilast (N=xxx) <sup>b</sup> |
| xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | ××× | Placebo<br>(N=xxx) <sup>b</sup> |
| xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | ××× | Overall (N=xxx) <sup>b</sup> |

Source Program: xxxxxxxxsas

Adverse events coded with MedDRA Coding Dictionary Version XXX.

b The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall.

STATKING Clinical Services (month day, year)

Table 6. Number and Proportion of Patients with Treatment-Related Adverse Events STALICIA SA - Study No. STP1-C004
Safety Population (N=xxx)

Page x of y

| Adverse Event Category <sup>a,b</sup> : | STP1mg<br>ibudilast<br>(N=xxx)° | Xmg<br>last<br>xx)° | STP1-<br>ibud<br>(N=) | STP1mg ibudilast (N=xxx)° | Pla<br>(N=) | Placebo<br>(N=xxx)° | Ove<br>(N=) | Overall (N=xxx)° |
|---|---|---|---|---|---|---|---|---|
| Total Number of Treatment-Related Adverse Events (AEs) | ××× | ^ | ××× | × | × | XXX | × | ××× |
| Patients with at Least One Treatment-Related AE | xxx (xxx) | (xx) | xxx (xxx) | (xxx) | ××× | (xxx) | ××× | xxx (xxx) |
| System Organ Class 1 | XXX ( | (xxx) | ××× | (xxx) | ××× | (XXX) | ××× | (xxx) |
| Preferred Term 1 | xxx ( | (xxx) | ××× | (xxx) | ××× | (xxx) | ××× | xxx (xxx) |
| Preferred Term 2 | XXX () | (xxx) | ××× | (xxx) | ××× | (xxx) | XXX | xxx (xxx) |
| System Organ Class 2 | XXX (; | (XXX) | ××× | (XXX) | ××× | (xxx) | ××× | (xxx) |
| Preferred Term 1 | xxx (; | (xxx) | xxx (xxx) | (xxx) | ××× | (xxx) | ××× | xxx (xxx) |
| Preferred Term 2 | xxx (xxx) | (XX) | xxx (xxx) | (000) | XXX (XXX) | ( ××× ) | XXX (XXX) | 1000) |


b A treatment-related AE is any AE with a relationship to study drug of Related.
c The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall.
STARKING Clinical Services (month day, year)

Source Program: xxxxxxx.sas

Table 7. Number and Proportion of Patients with Treatment-Related Adverse Events that Led to Study Drug
Discontinuation
STALICIA SA - Study No. STP1-C004
Safety Population (N=xxx) Page x of y

| Adverse Event Category <sup>a,b</sup> : | STP1-\mng ibudilast (N=xxx)° | STP1-\_mg ibudilast (N=xxx)° | Placebo<br>(N=xxx)° | Overall (N=xxx)° |
|---|---|---|---|---|
| Total Number of Treatment-Related Adverse Events (AEs) that Led to Study Drug Discontinuation | ××× | ×× | ×<br>×<br>× | ×<br>×<br>× |
| Patients with at Least One Treatment-Related AE that Led to Study Drug Discontinuation | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| System Organ Class 1 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 1 | XXX (XXX) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 2 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| System Organ Class 2 | XXX (XXX) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 1 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 2 | xxx (xxx) | xxx (xxx) | vvv (vvv) | vvv (vvv) |


b A treatment-related AE is any AE with a relationship to study drug of Related.
c The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall.
STATKING Clinical Services (month day, year)
Source Program: xxxxxxxx.sas

Table 8. Number and Proportion of Patients with Serious Adverse Events STALICIA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

Adverse Event Categorya: Total Number of Serious Adverse Events (SAEs) Patients with at Least One SAE System Organ Class 1 Preferred Term 2 Preferred Term 1 STP1-Xmg ibudilast (N=xxx)<sup>b</sup> xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) XXX STP1-\\_mg
ibudilast
(N=xxx)<sup>b</sup> xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) ××× xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) Placebo (N=xxx)<sup>b</sup> XXX xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) Overall (N=xxx) b XXX

System Organ Class 2

Preferred Term 2 Preferred Term 1

xxx (xxx)

xxx (xxx) xxx (xxx) xxx (xxx)

xxx (xxx) xxx (xxx)

xxx (xxx)

xxx (xxx) xxx (xxx)

xxx (xxx)

xxx (xxx) xxx (xxx)

<sup>b</sup> The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall. STATKING Clinical Services (month day, year) Adverse events coded with MedDRA Coding Dictionary Version XXX.

Source Program: xxxxxxx.sas


Table 9. Number and Proportion of Patients with Treatment-Related Serious Adverse Events STALICIA SA - Study No. STP1-C004
Safety Population (N=xxx)

Page x of y

| Adverse Event Category <sup>a,b</sup> : | STP1-Xng ibudilast (N=xxx)° | STP1-Xng ibudilast (N=xxx)° | Placebo<br>(N=xxx)° | Overall (N=xxx)° |
|---|---|---|---|---|
| Total Number of Treatment-Related Serious Adverse Events (SAEs) | ××× | ××× | ××× | ××× |
| Patients with at Least One Treatment-Related<br>SAE | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| System Organ Class 1 | xxx (xxx) | xxx (xxx) | xxx (xxx) | XXX (XXX) |
| Preferred Term 1 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 2 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| System Organ Class 2 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 1 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 2 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |


b A treatment-related AE is any AE with a relationship to study drug of Related.
c The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall.
STARKING Clinical Services (month day, year)

Source Program: xxxxxxx.sas

Table 10. Number and Proportion of Patients with Treatment-Related Serious Adverse Events that Led to Study Drug Discontinuation STALICLA SA - Study No. STP1-C004

Page x of y

Safety Population (N=xxx)

| System Organ Class 2 Preferred Term 1 Preferred Term 2 | System Organ Class 1 Preferred Term 1 Preferred Term 2 | Patients with at Least One Treatment-Related SAE that Led to Study Drug Discontinuation | Total Number of Treatment-Related Serious Adverse Events (SAEs) that Led to Study Drug Discontinuation | Adverse Event Category <sup>a,b</sup> : |
|---|---|---|---|---|
| × × ×<br>× × × | × | ××× | | STI<br>ibu |
| (xxx)<br>(xxx) | xxx (xxx)<br>xxx (xxx) | xxx (xxx) | ××× | STP1-\_mg ibudilast (N=xxx)° |
| XXX ( | × | xxx (xxx) | ××× | STP1-\_mg ibudilast (N=xxx)° |
| (xxx)<br>(xxx) | (xxx)<br>(xxx) | xxx) | × | rP1-\_mg<br>budilast<br>(N=xxx)° |
| × × ×<br>× × × | × × ×<br>× × × | ××× | × | P1a |
| ( | (xxx)<br>(xxx) | (xxx) | ××× | Placebo<br>(N=xxx)° |
| * * * | × × ×<br>× × × | ××× | × | Ove<br>(N=: |
| xxx (xxx)<br>xxx (xxx) | xxx (xxx)<br>xxx (xxx) | xxx (xxx) | ××× | Overall (N=xxx)° |


b A treatment-related AE is any AE with a relationship to study drug of Related.
c The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall.
STARKING Clinical Services (month day, year)

Source Program: xxxxxxx.sas

Table 11. Number and Proportion of Patients with Adverse Events of Special Interest STALICIA SA - Study No. STP1-C004
Safety Population (N=xxx)

Page x of y

| Adverse Event Category®: | STP1mg ibudilast (N=xxx) <sup>b</sup> | STP1ng ibudilast (N=xxx) <sup>b</sup> | Placebo<br>(N=xxx) <sup>b</sup> | Overall (N=xxx) <sup>b</sup> |
|---|---|---|---|---|
| Total Number of Adverse Events of Special Interest (AESIs) | ××× | ××× | ××× | ××× |
| Patients with at Least One AESI | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| System Organ Class 1 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (; |
| Preferred Term 1 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (z |
| Preferred Term 2 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| System Organ Class 2 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 1 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 2 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx |


b The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall. STATKING Clinical Services (month day, year)
Source Program: xxxxxxxx.sas

Table 12. Number and Proportion of Patients with Adverse Events of Special Interest that Led to Study
Drug Discontinuation
STALICIA SA - Study No. STP1-C004
Safety Population (N=xxx)

Page x of y

| STP1-Xng STP1-Xng Ibudilast Placebo Overall (N=xxx)b (N=xxx)b (N=xxx)b (N=xxx)b xxx xxx xxx xxx x | System Organ Class 2 Preferred Term 1 Preferred Term 2 | System Organ Class 1 Preferred Term 1 Preferred Term 2 | Total Number of Adverse Events of Special Interest (AESIs) that Led to Study Drug Discontinuation Patients with at Least One AESI that Led to Study Drug Discontinuation | Adverse Event Category®: |
|---|---|---|---|---|
| g STP1—Xng Placebo (N=xxx) b (N=xxx) b xxx (xxx) xxx (xxx) | × × × × × × | × × × × × | XXX | STP<br>ibu<br>(N |
| Placebo (N=xxx) b xxx xxx xxx (xxx) | ( | (xxx)<br>(xxx) | (xxx) | 1-\text{mg} dilast =xxx) b |
| xxxy) b (xxxx) | xxx (xxx)<br>xxx (xxx) | xxx (xxx)<br>xxx (xxx) | xxx (xxx) | STP1-\_mg ibudilast (N=xxx) <sup>b</sup> |
| | xxx () xxx () xxx () | | ××× () | Place<br>(N=xx |
| Overall (N=xxx) <sup>b</sup> xxx xxx xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) xxx (xxx) | (xx)<br>(xx) | (xxx) | (x<br>x<br>x | م (×<br>م (× |
| ixxx) b (xxx) | × × ×<br>× × × | × | ×<br>×<br>× | Ove |
| I I | ( | (xxx)<br>(xxx) | ( | erall<br>exxx) b |

Source Program: xxxxxxx.sas


b The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall.

STATKING Clinical Services (month day, year)

Table 13. Number and Proportion of Patients with Adverse Events by Relationship to Study Drug
STALICIA SA - Study No. STP1-C004
Safety Population (N=xxx)

Page x of y

| | $srp1-\underset{(N=xxx)^b}{\longrightarrow} mg ibudilast$ | mg ibudilast<br>(N=xxx) <sup>b</sup> | STP1-\_mg ibudilast (N=xxx) <sup>b</sup> | ibudilast<br>xx) <sup>b</sup> | Placebo<br>(N=xxx) <sup>b</sup> | ebo<br>xx) b |
|---|---|---|---|---|---|---|
| Adverse Event Categoryª: | Not Related | Related | Not Related | Related | Not Related | Related |
| Total Number of Adverse Events (AEs) | ××× | ××× | ××× | ××× | ××× | ××× |
| Patients with at Least One AE | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| System Organ Class 1 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 1 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 2 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| System Organ Class 2 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 1 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 2 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |


b The denominator for all proportions is the number of Safety population patients in the corresponding treatment group. STATKING Clinical Services (month day, year)
Source Program: xxxxxxxx.sas

Table 14. Number and Proportion of Patients with Adverse Events by Severity STALICLA SA - Study No. STP1-C004
Safety Population (N=xxx)

Page x of y

| | STP | STP1- $\times$ mg ibudilast (N=xxx) <sup>b</sup> | last | STP1 | $STP1-$ ng ibudilast $(N=xxx)^b$ | ilast | | Placebo<br>(N=xxx) <sup>b</sup> | |
|---|---|---|---|---|---|---|---|---|---|
| Adverse Event Categorya: | Mild | Moderate | Severe | Mild | Moderate | Severe | Mild | Moderate | Severe |
| Total Number of Adverse Events (AEs) | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× |
| Patients with at Least One AE | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| System Organ Class 1 | (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 1 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 2 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| System Organ Class 2 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 1 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 2 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |


b The denominator for all proportions is the number of Safety population patients in the corresponding treatment group. STATKING Clinical Services (month day, year)
Source Program: xxxxxxxx.sas

Table 15. Vital Sign Parameter Summary Statistics STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| Treatment | STP1-Xmg<br>ibudilast | | | | | STP1mg | | | | | Placebo | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter<br>(units) <sup>a</sup> | (xxx) | | | | | (xxx) | | | | | (xxx)<br>(xxx | | | | |
| Visit | Baseline | XXXXXX | | ×××××× | | Baseline | ××××× | | XXXXXX | | Baseline | XXXXXX | | ××××× | |
| Time | ××× | XXXX | ×××× | xxxx | XXXX | ×××× | ×××× | ×××× | XXXX | ×××× | ×××× | XXXX | ×××× | ×××× | XXXX |
| Data<br>Type <sup>b</sup> | RAW | RAW | CFB | RAW | CFB | RAW | RAW | CFB | RAW | CFB | RAW | RAW | CFB | RAW | CFB |
| n | ××× | ××× | ××× | ××× | XXX | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× |
| Mean | XXX | XXX | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× |
| Std Dev | ××× | XXX | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× |
| Median | ××× | XXX | ××× | ××× | XXX | ××× | ××× | ××× | XXX | ××× | ××× | ××× | ××× | ××× | ××× |
| Min | ××× | XXX | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× |
| Max | ××× | ××× | ××× | ××× | XXX | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× |

Vital sign parameters in this table include temperature and respiratory rate.

b RAW = observed data recorded in database; CFB = change from baseline = (results at current visit) - (Baseline results).

STATKING Clinical Services (month day, year)

Source Program: xxxxxxx.sas


Table 16. Orthostatic Vital Sign Parameter Summary Statistics STALICIA SA - Study No. STP1-C004
Safety Population (N=xxx)

Page x of y

| | rla cebo | | STP1ng<br>ibudilast | ibudilast | Treatment |
|---|---|---|---|---|---|
| | (xxx)<br>(xxx) | | (xxx)<br>(xxx) | ( xxx) xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Parameter (units) <sup>a</sup> |
| xxxxxx | baseline | XXXXXX | Baseline<br>xxxxxx | Baseline xxxxxx | Visit |
| × | × | ×××× | × | × | Time |
| RAW<br>CFB | RAW<br>CFB | RAW<br>CFB | CFB<br>RAW<br>RAW<br>CFB | RAW<br>CFB<br>CFB | Data<br>Type <sup>b</sup> |
| × ×<br>× × | × × × × × | × × × × | × | × ×× ×<br>× ×× × | n |
| ××× | × × × × × × | ×××<br>××× | × | × ×× ×<br>× ×× × | Mean |
| ××× | × × × × × × | XXX<br>XXX | × | × ×× ×<br>× ×× × | Std Dev |
| × ×<br>× × | × × × × × | × × × | × | × | Median |
| ×××<br>××× | × × × × × × | ×××<br>××× | × | × × × × × × | Min |
| × × × × × | × × × × × × | ×××<br>××× | × × × × × × × | × ×× ×<br>× ×× × | Max |

Vital sign parameters in this table include orthostatic heart rate, orthostatic diastolic blood pressure, and orthostatic systolic blood pressure taken in the supine position.

b RAW = observed data recorded in database; CFB = change from baseline = (results at current visit) - (Baseline results).

STATKING Clinical Services (month day, year)

Source Program: xxxxxxx.sas

Table 17.

Page x of y

| Overall | | Placebo | STP1ng | Treatment STP1-Xmg ibudilast | |
|---|---|---|---|---|---|
| (xxx) | (xxx) | ××××××××××××××××××××××××××××××××××××××× | (xxx)<br>(xxxxxxxxx | (units) xxxxxxxxx (xxx) | Parameter |
| Baseline xxxxxx xxxxxx | XXXXXX<br>XXXXX | xxxxxx<br>Baseline | xxxxxx<br>Baseline | Visit <sup>a</sup> Baseline xxxxx | |
| ×× ×× ×<br>×× ×× × | × | × | × | Time xxxx xxxx | |
| RAW<br>CFB<br>CFB | RAW<br>CFB<br>RAW<br>CFB | RAW<br>CFB<br>RAW | RAW<br>CFB<br>RAW<br>RAW<br>CFB | Type <sup>b</sup> RAW RAW CFB | Data |
| ** ** * | × | × ××<br>× ×× | × | x x x x x x x x x x x x x x x x x x x | |
| ** * * * | × | × | * * * * * * | Mean xxx xxx | |
| ** ** * | × | × ××<br>× ×× | * * * * * * | Std Dev | |
| ** * * * | × | × | * * * * * * | Median xxx xxx xxx | : |
| ** ** * | × | × | ** * * * | xxxx xx | |
| ** ** ** | × | × ××<br>× ×× | * * * * * * | X X X X X X X X X X X X X X X X X X X | |

The baseline raw value for each parameter is calculated using the average of the triplicate values from the ECG performed on Day 1 pre-dose.

b Raw = observed data; CFB = change from baseline = (results at current visit) - (Baseline results).

STARKING Clinical Services (DDMMMYYYYY)


Source Program: xxxxxxx.sas

Table 18. ECG Results Shift Table by Visit and Clinical Significance STALICIA SA - Study No. STP1-C004
Safety Population (N=xxx)

Page x of y

Baselineª/Visitb,c

| Overall | Placebo | STP1ng<br>ibudilast | STP1ng<br>ibudilast | Treatment |
|---|---|---|---|---|
| × | × | × | ×××××<br>×××××××××××××××××××××××××××××××× | Visit |
| xxx (xx)<br>xxx (xx) | xxx (xx)<br>xxx (xx) | XXX (XX) XXX (XX) | XXX (XX) XXX (XX) | Normal/ |
| xxx (xx)<br>xxx (xx) | (xx) xxx (xx) xxx (xx) | xxx (xx)<br>xxx (xx) | XXX (XX) XXX (XX) | Normal/<br>Abnormal<br>CS |
| (xx) xxx (xx) xxx (xx) | xxx (xx)<br>xxx (xx) | xxx (xx) xxx (xx) | ××× (××) ××× (××) | Normal/<br>Abnormal |
| (xx) xxx (xx) xxx (xx) | xxx (xx)<br>xxx (xx)<br>xxx (xx) | xxx (xx) xxx (xx) | ××× (××) ××× (××) | Abnormal<br>CS/<br>Normal |
| xxx (xx) xxx (xx) | xxx (xx)<br>xxx (xx) | xxx (xx)<br>xxx (xx) | ××× (××) ××× | Abnormal<br>CS/<br>Abnormal CS |
| xxx (xx)<br>xxx (xx) | xxx (xx)<br>xxx (xx) | xxx (xx)<br>xxx (xx) | xxx (xx)<br>xxx (xx) | Abnormal CS/ |
| xxx (xx) xxx (xx) | xxx (xx)<br>xxx (xx) | (xx) xxx (xx) xxx (xx) | ××× (××) ××× (××) | Abnormal / NCS/ |
| xxx (xx)<br>xxx (xx) | XXX (XX)<br>XXX (XX) | (xx) xxx (xx) xxx (xx) | ××× (××) ××× (××) | Abnormal<br>NCS/<br>Abnormal<br>CS |
| XXX (XX) XXX (XX) | xxx (xx)<br>xxx (xx) | xxx (xx) xxx (xx) | xxx (xx)<br>xxx (xx) | Abnormal<br>NCS/<br>Abnormal NCS |

Source Program: xxxxxxx.sas


The baseline ECG result performed in triplicate is determined as outlined in section 4.2 of the SAP.

b A normal result are those results that the Principal Investigator determined to be within normal range. CS = Clinically Significant.

NCS= Not Clinically Significant.

c The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall.

STATKING Clinical Services (month day, year)

Table 19. ECG Results Shift Table by Visit STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

Baselinea/Visitb,c

| Treatment | Parameter | Visit | Normal/Normal | Normal/Normal Normal/Abnormal Abnormal/Normal Abnormal/Abnormal | Abnormal/Normal | Abnormal/Abno |
|---|---|---|---|---|---|---|
| STP1- mg ibudilast | ××××× | xxxxx | xxx (xxxx) | xxx (xxxx) | xxx (xxxx) | xxx (xxxx) |
| ı | | ××××× | xxx (xxxx) | xxx (xxxx) | xxx (xxxx) | xxx (xxxx) |
| STP1- mg ibudilast | ××××× | ××××× | xxx (xxxx) | xxx (xxxx) | xxx (xxxx) | xxx (xxxx) |
| Î | | XXXXXX | xxx (xxxx) | xxx (xxxx) | xxx (xxxx) | xxx (xxxx) |
| Placebo | ××××× | XXXXXX | xxx (xxxx) | xxx (xxxx) | xxx (xxxx) | xxx (xxxx) |
| | | XXXXXX | xxx (xxxx) | xxx (xxxx) | xxx (xxxx) | xxx (xxxx) |
| Overall | ××××× | XXXXXX | xxx (xxxx) | xxx (xxxx) | xxx (xxxx) | xxx (xxxx) |
| | | XXXXXX | xxxx (xxxx) | xxx (xxxx) | xxx (xxxx) | xxx (xxxx) |

Parameters in this table are T wave, U wave and ECG Interpretation.

The baseline ECG result performed in triplicate is determined as outlined in section 4.2 of the SAP.

b A normal result are those results that the Principal Investigator determined to be within normal range.

c The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall. STATKING Clinical Services (DDMMMYYYY)

Source Program: xxxxxxxx.sas

Table 20. Blood Chemistry Parameter Summary Statistics STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| | | Overall | | Placebo | | ibudilast | STP1-Xmg | | TRUCTTASC | STP1-Xmg | Treatment |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | (xxx) | XXXXXXXXXXX | ĺ | (xxx)<br>(xxx) | | (xxx) | ××××××××××××××××××××××××××××××××××××××× | | (×××) | ×××××××××××××××××××××××××××××××××××××× | Parameter (units) |
| ×××××<br>××××× | XXXXXX | xxxxxx | × | Baseline | × ×<br>× ×<br>× ×<br>× × | × | Baseline | ×××××<br>×××××× | ***** | Baseline | Visit |
| RAW<br>CFB | RAW<br>CFB | CFB<br>RAW | RAW<br>CFB<br>RAW | RAW | RAW | RAW<br>CFB | RAW | RAW | RAW<br>CFB | RAW | Data<br>Type <sup>a</sup> |
| × ×<br>× × | × ×<br>× × | × ×<br>× × | × | ××× | × ×<br>× × | × ×<br>× × | ××× | × ×<br>× × | × × × | ××× | n |
| × ×<br>× × | × ×<br>× × | × ×<br>× × | × ×× | ××× | × ×<br>× ×<br>× × | × ×<br>× × | ××× | × ×<br>× × | × ×<br>× × | ××× | Mean |
| × ×<br>× × | × ×<br>× × | × ×<br>× × | × ××<br>× ×× | ××× | × ×<br>× ×<br>× × | × ×<br>× × | XXX | × ×<br>× × | ×××<br>××× | ××× | Std Dev |
| × ×<br>× × | × × × × | × ×<br>× × | × ××<br>× ×× | ××× | × ×<br>× × | × ×<br>× × | XXX | × ×<br>× × | ×××<br>××× | ×<br>×<br>× | Median |
| × ×<br>× × | × × × × | × ×<br>× × | × ××<br>× ×× | ××× | × ×<br>× × | × ×<br>× × | ××× | × ×<br>× × | × × × × × | ××× | Min |
| × ×<br>× × | × ×<br>× × | × ×<br>× × | × ××<br>× ×× | ××× | × ×<br>× ×<br>× × | × ×<br>× × | ××× | × ×<br>× × | ×××<br>××× | ××× | Max |

RAW = observed data recorded in database; CFB = change from baseline = (results at current visit) - (Baseline results). STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Table format will be repeated for Hematology, Coagulation and Urinalysis.


Table 24. Summary of Qualitative Urinalysis Results by Parameter

Page x of y

| Safety Pop | STALICIA SA - | |
|---------------------------|---------------------------------|---|
| Safety Population (N=xxx) | ALICLA SA - Study No. STP1-C004 | 1 |

| Parameter | Visit | Result | STP1mg ibudilast (N=xxx) <sup>a</sup> | STP1mg ibudilast (N=xxx) a | Placebo<br>(N=xxx) a | Overall (N=xxx) a |
|---|---|---|---|---|---|---|
| XXXXX | ×××× | ×××××× | xxx (xxx) | xxx (xxx) | xxx (xxx) | × |
| | | XXXXXX | xxx (xxx) | xxx (xxx) | xxx (xxx) | ×× |
| | | ×××××× | xxx (xxx) | | xxx (xxx) | xxx (xxx) |
| | ×××× | ×××××× | | | | × |
| | | XXXXXX | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx |
| | | XXXXXX | | _ | _ | ×× |

The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall. STATKING Clinical Services (DDMMMYYYY)
Source Program: xxxxxxx.sas


Table 25. Blood Chemistry Results Shift Table by Visit and Clinical Significance STALICIA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| (xxx) (xxx) | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Parameter (units) |
|---|---|---|---|
| ××××××××××××××××××××××××××××××××××××××× | Placebo Overall | STP1mg ibudilast STP1mg ibudilast | Treatment |
| × | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | X X X X X X X X X X X X X X X X X X X | Visit |
| × | XXX (XX) XXX (XX) XXX (XX) XXX (XX) XXX (XX) | XXX (XX) XXX (XXX) XXX (XXX) XXX (XXXX (XXX (XXXX (XXX (XXXX (XXX (XXXX (XXX (XX (XXX (XX (X ( | Normal/ |
| ××× (××) (××) | XXX (XX) XXX (XX) XXX (XX) XXX (XX) | XXX (XX) XXX (XX) XXX (XX) | Normal/<br>Abnormal |
| ××× ×× (××) | (xx) xxx (xx) xx (xx) | XXX (XX) XXX (XX) XXX (XX) XXX (XX) | Normal/<br>Abnormal |
| ××× ×× (××) | XXX (XX) XXX (XX) XXX (XX) | XXX (XX) XXX (XX) XXX (XX) | Abnormal CS/ |
| ××× (××) ××× (××) | XXX XXX (XXX) (XXX) (XXX) | XXX (XX) XXX (XX) XXX (XX) XXX (XX) | Baseline/Visita,b Abnormal Al CS/ Abnormal Al CS CS |
| ××× ×× (×× ×× | XXX (XX) XXX (XX) XXX (XX) XXX (XX) | XXX XX | Abnormal CS/ Abnormal NCS |
| ××× ×× (×× ×× | XXX (XX) XXX (XX) XXX (XX) XXX (XX) | XXX XX | Abnormal<br>NCS/<br>Normal |
| ××× ×× (×× ×× | XXX (XX) XXX (XX) XXX (XX) XXX (XX) | XXX XX | Abnormal<br>NCS/<br>Abnormal |
| × | (xx)<br>(xx)<br>(xx)<br>(xx)<br>(xx)<br>(xx) | XXX (XX) XXX (XX) XXX (XX) | Abnormal<br>NCS/<br>Abnormal |


A normal result are those results that the Principal Investigator determined to be within normal range. CS = Clinically Significant.

NCS= Not Clinically Significant.

b The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall.

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Table format will be repeated for Hematology, Coagulation, Urinalysis, and Blood Chemistry Results for Electrolytes Laboratory parameters in Table 25 will exclude sodium, chloride, calcium, magnesium, phosphate, and potassium. Laboratory parameters in Table 29 will include sodium, chloride, calcium, magnesium, phosphate, and potassium.

Table 30. Blood Chemistry Results for Electrolytes Shift Table by Visit and Range of Normal Results STALICIA SA - Study No. STP1-C004
Safety Population (N=xxx)

Page x of y

| | Laboratory Parameter (units) | (***) | ĺ | | | | | | (xxx) | (999) |
|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment | STP1-Xmg<br>ibudilast | | STP1-\_mg | | Placebo | | Overall | xxxxxxxx | |
| | Visit | XXXXXX | × | xxxxxx | ***** | × | XXXXXX | × | ×××××× | ×××××<br>×××××× |
| | High/<br>High | xxx (xx) | (xx) xxx (xx) | xxx (xx) | xxx (xx) | ××× (××) | _ | XXX (XX)<br>XXX (XX) | xxx (xx) | XXX (XX) |
| | High/<br>Normal | xxx (xx) | xxx (xx) | xxx (xx) | xxx (xx) | XXX (XX) | _ | XXX (XX)<br>XXX (XX) | xxx (xx) | XXX (XX) |
| | High/<br>Low | xxx (xx) | xxx (xx) | xxx (xx) | xxx (xx) | XXX (XX) | _ | XXX (XX)<br>XXX (XX) | xxx (xx) | XXX (XX) |
| Ba | Normal/<br>High | xxx (xx) | xxx (xx)<br>xxx (xx) | xxx (xx) | xxx (xx) | ××× (××) | _ | xxx (xx)<br>xxx (xx) | xxx (xx) | XXX (XX) |
| Baseline/Visita,b | Normal/<br>Normal | xxx (xx) | xxx (xx)<br>xxx (xx) | xxx (xx) | xxx (xx) | xxx (xx) | _ | XXX (XX)<br>XXX (XX) | xxx (xx) | XXX (XX) |
| ta,b | Normal/<br>Low | xxx (xx) | xxx (xx)<br>xxx (xx) | xxx (xx) | xxx (xx) | ××× (××) | XXX (XX) | XXX (XX)<br>XXX (XX) | xxx (xx) | XXX (XX) |
| | Low/<br>High | xxx (xx) | XXX (XX) | xxx (xx) | xxx (xx)<br>xxx (xx) | ××× (××) | XXX (XX) | XXX (XX)<br>XXX (XX) | xxx (xx) | XXX (XX) |
| | Low/<br>Normal | xxx (xx) | XXX (XX) | xxx (xx) | xxx (xx) | ×××<br>×××<br>(××) | XXX (XX) | XXX (XX)<br>XXX (XX) | xxx (xx) | XXX (XX) |
| | Low/ | xxx (xx) | xxx (xx)<br>xxx (xx) | xxx (xx) | xxx (xx) | ××× (××) | XXX (XX) | ××× (××) ××× (××) | xxx (xx) | xxx (xx)<br>xxx (xx) |

Laboratory parameters include: sodium, chloride, calcium, magnesium, phosphate, and potassium.


A normal result are those results that the Principal Investigator determined to be within normal range.

b The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall.

STATKING Clinical Services (month day, year)

Source Program: xxxxxxx.sas

Table 31. Number and Proportion of Patients with Blood Chemistry Results for Electrolytes Outside of
Normal Range
STALICLA SA - Study No. STP1-C004
Safety Population (N=xxx)

Page x of y

| | 17.<br>0 | J<br>)<br>:<br>:<br>t | STP1mg ibudilast | STP1-\_mg ibudilast | Placebo |
|---|---|---|---|---|---|
| Parameter (units) | Visit | Result | (N=xxx) a | (N=xxx) a | (N=XXX) a |
| xxxxxxxxx (xxx) | xxxxxx | Low | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| | | High | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| | xxxxxx | Low | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| | | High | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| xxxxxxxxxx (xxx) | ××××× | Low | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| | | High | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| | XXXXXX | Low | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| | | High | xxx (xxx) | 000 (000) | xxx (xxx) |

Source Program: xxxxxxx.sas The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall. STATKING Clinical Services (DDMMMYYYY)

Laboratory parameters include: sodium, chloride, calcium, magnesium, phosphate, and potassium.


Table 32. Summary Statistics of Ibudilast and Bumetanide Plasma Concentration Levels by Treatment, Visit and Time

STALICIA SA - Study No. STP1-C004

PK Population (N=xxxx)

Page x of y

| | | | | | | | Bumetanide | | | | | | | | Ibudilast | Drug <sup>a</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | STP1\\ng ibudilast | | | | STP1 mg ibudilast | | | | STP1-Xmg ibudilast | | | | STP1 mg ibudilast | Treatment |
| | ××× | | ××× | | ××× | | ××× | | ××× | | ××× | | ××× | | ××× | Visit |
| XXX | XXX | ××× | XXX | ××× | XXX | ××× | ××× | ××× | XXX | ××× | ××× | ××× | XXX | ××× | ××× | Time (hrs) |
| XXX | ××× | ×× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | n |
| XXX | ××× | ×× | ××× | ××× | ××× | ××× | ×× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | Mean |
| ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | XXX | ××× | ××× | ××× | ××× | ××× | ××× | Std Dev |
| ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | Median |
| XXX | ××× | ×× | ××× | ××× | ××× | ××× | ××× | ××× | ×× | ××× | ×× | ××× | ××× | ××× | ××× | Min |
| ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | Max |

Concentration levels measured in units of xxx. STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Table 33. Summary Statistics of Ibudilast and Bumetanide Urine Concentration Levels by Treatment, Visit and Time STALICLA SA - Study No. STP1-C004 PK Population (N=xxx)

Page x of y

| | | | Bumetanide | | | | Ibudilast | Drugª |
|---|---|---|---|---|---|---|---|---|
| | STP1 ng ibudilast | | STP1 mg ibudilast | | STP1 mg ibudilast | | STP1 mg ibudilast | Treatment |
| ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | Visit |
| × ×<br>× × | × × × × × × | × ×<br>× × | × ×<br>× × | × ×<br>× × | × × × × × | × ×<br>× × | X X X | Time (hrs) |
| × × | × × | × × | × × | × × | × × | × × | × × | p |
| × × | × × | × × | × × | × × | × × | × × | × × | |
| × × | × × | × × | × × | × × | × × | × × | × × | Mean |
| × × | × × | × × | × × | × × | × × | × × | × × | |
| × × | × × | × × | × × | × × | × × | × × | × × | Std Dev |
| × × | × × | × × | × × | × × | × × | × × | × × | |
| × × | × × | × × | × × | × × | × × | × × | × × | Median |
| × × | × × | × × | × × | × × | × × | × × | × × | |
| × × | × × | × × | × × | × × | × × | × × | × × | Min |
| × × | × × | × × | × × | × × | × × | × × | × × | |
| × × | × × | × × | × × | × × | × × | × × | × × | Max |
| × × | × × | × × | × × | × × | × × | × × | × × | |

Concentration levels measured in units of xxx. STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Table 34. Summary Statistics of Estimated PK Plasma Parameters for Ibudilast by Treatment STALICIA SA - Study No. STP1-C004
PK Population (N=xxx)

Page x of y

Part 1 of 2: STP1- 📉 ibudilast

| | | Overall | | | | | | | | | Day 14 | | | | | | | | Day 1 | Visit | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ARcmax | ARauc | AUC <sub>0-*</sub> (hrs* xxx/mL) | Cl/F (mL/hrs) | Vz/F (mL) | AUC0-last (hrs* xxx/mL) | AUC0-12h,ss (hrs* xxx/mL) | AUC0-tau(6h),ss (hrs* xxx/mL) | t <sub>1/2</sub> (hrs) | Ctrough (XXX /mL) | Tmax (hrs) | Cmax,ss (xxx /mL) | Cl/F (mL/hrs) | Vz/F (mL) | AUC0-last (hrs* xxx/mL) | AUC0-tau(6h), Day 1 (hrs* xxx/mL) | t <sub>1/2</sub> (hrs) | Ctrough (XXX /mL) | Tmax (hrs) | Cmax, Day 1 (XXX/mL) | Parameter (units) | |
| ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | XXX | ××× | ××× | ××× | ××× | XXX | ××× | ××× | ××× | ××× | n | |
| ××× | ××× | ××× | ××× | ××× | XXX | ××× | ××× | ××× | XXX | XXX | ××× | ××× | ××× | ××× | XXX | ××× | ××× | ××× | ××× | Mean | |
| ××× | XXX | ××× | ××× | XXX | XXX | XXX | xxx | ××× | XXX | XXX | ××× | ××× | ××× | ××× | XXX | XXX | xxx | XXX | ××× | Std Dev | |
| ××× | ××× | ××× | XXX | ××× | ××× | ××× | ××× | ××× | ××× | XXX | ××× | ××× | ××× | ××× | XXX | ××× | ××× | ××× | ××× | CV% | |
| ××× | ××× | ××× | ××× | ××× | XXX | ××× | XXX | ××× | XXX | XXX | ××× | ××× | XXX | ××× | XXX | ××× | XXX | ××× | ××× | Mean | Geometric |
| ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× | XXX | ××× | ××× | ××× | ××× | XXX | ××× | ××× | ××× | ××× | 90% CI | Lower |
| ××× | XXX | ××× | ××× | ××× | XXX | ××× | XXX | XXX | XXX | XXX | ××× | ××× | ××× | ××× | XXX | ××× | XXX | ××× | ××× | 90% CI | Upper |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Table 34. Summary Statistics of Estimated PK Plasma Parameters for Ibudilast by Treatment STALICIA SA - Study No. STP1-C004
PK Population (N=xxx)

Page x of y

Part 2 of 2: STP1- mg ibudilast

| , |
|---|

| Overall | Day 14 | | Visit Day 1 |
|---|---|---|---|
| AUCo-= (hrs* xxx/mL)<br>ARauc<br>ARcmax | Cmax.ss(XXX/mL) Tmax (hrs) Ctrough (xxx /mL) tl/2 (hrs) AUCo-tau(6h),ss (hrs* xxx/mL) AUCo-tast (hrs* xxx/mL) Vz/F (mL) C1/F (mL/hrs) | Tmax (hrs) Ctrough (xxx /mL) t1/2 (hrs) AUCo-tau (sh), Day 1 (hrs* xxx/mL) AUCo-taust (hrs* xxx/mL) Vz/F (mL) C1/F (mL/hrs) | Parameter (units) Cmax,Day 1 (xxx/mL) |
| × × ×<br>× × × | | * | n |
| × × ×<br>× × × | * | * | Mean |
| × × ×<br>× × × | * | * | Std Dev |
| × | * | * | CV% |
| × × ×<br>× × × | | * | Geometric<br>Mean |
| × × ×<br>× × × | * | * | Lower<br>90% CI |
| × × ×<br>× × × | * | * | Upper<br>90% CI<br>xxx |

STATKING Clinical Services (month day, year) Source Program: xxxxxxxx.sas

Table 35. Summary Statistics of Estimated PK Plasma Parameters for Bumetanide by Treatment STALICIA SA - Study No. STP1-C004
PK Population (N=xxx)

Page x of y

Part 1 of 2: STP1-Xmg ibudilast

| Overall | Day 1 Day 14 | Visit |
|---|---|---|
| Call | 14 | ř.<br>t |
| AUCo (hrs* xxx/mL)<br>ARauc<br>ARcmax | Cmax,Day 1 (XXX/mL) Tmax (hrs) Ctrough (XXX /mL) t1/2 (hrs) AUCo-tau (6h),Day 1 (hrs* xxx/mL) AUCo-tast (hrs* xxx/mL) VZ/F (mL/hrs) C1/F (mL/hrs) Cmax,ss (XXX /mL) Tmax (hrs) Ctrough (XXX /mL) t1/2 (hrs) AUCo-tau (6h),Ss (hrs* xxx/mL) AUCo-tau (6h),Ss (hrs* xxx/mL) AUCo-12h,ss (hrs* xxx/mL) AUCo-12h,ss (hrs* xxx/mL) C1/F (mL/hrs) C1/F (mL/hrs) | Parameter (units) |
| × × ×<br>× × × | | n |
| × × ×<br>× × × | | Mean |
| × × ×<br>× × × | | Std Dev |
| × × ×<br>× × × | | CV% |
| × × ×<br>× × × | | Geometric<br>Mean |
| × × ×<br>× × × | | Lower<br>90% CI |
| × × ×<br>× × × | | Upper<br>90% CI |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas


Table 35. Summary Statistics of Estimated PK Plasma Parameters for Bumetanide by Treatment STALICIA SA - Study No. STP1-C004
PK Population (N=xxx)

Page x of y

Part 2 of 2: STP1- mg ibudilast

| | | | | | 1 |
|---|---|---|---|---|---|
| Overall | | | Day 14 | | Visit<br>Day 1 |
| AUCo-= (hrs* xxx/mL) ARauc ARcmax | AUCo-12h,ss (hrs* xxx/mL) AUCo-12at (hrs* xxx/mL) Vz/F (mL) Cl/F (mL/hrs) | Thax (DTS) Ctrough (XXX /ML) ti/2 (hTS) AUC0-tau(6h),ss (hTS* XXX/ML) | Vz/F (mL) Cl/F (mL/hrs) Cmax,ss (xxx /mL) | Tmax (hrs) Ctrough (xxx /mL) Ctrough (xxx /mL) ti/2 (hrs) AUCo-tau (6h), Day 1 (hrs* xxx/mL) AUCo-tast (hrs* xxx/mL) | Parameter (units) Cmax,Day 1 (xxx/mL) |
| × × × | × × × ×<br>× × × × | × | | × | n |
| × × × | × × × ×<br>× × × × | × | × ×× | × | Mean |
| × × × × i | × × × ×<br>× × × × | × × × × × × | | × | Std Dev |
| × × × | × | × | × × × × | × | CV% |
| × × × × · · | × × × ×<br>× × × × | × | : | × | Geometric<br>Mean |
| × × × ; | × × × ×<br>× × × × | × | X | × | Lower<br>90% CI |
| × × × : | × × × ×<br>× × × × | × | X | × | Upper<br>90% CI |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas


Table 36. Summary Statistics of Estimated PK Urine Parameters for Ibudilast by Treatment STALICIA SA - Study No. STP1-C004
PK Population (N=xxx)

Page x of y

Part 1 of 2: STP1-Xmg ibudilast

| Visit | Parameter | n | Mean | Std Dev | CV% | Geometric<br>Mean | Lower<br>90% CI | Upper<br>90% C |
|---|---|---|---|---|---|---|---|---|
| Day 1 | Excretion Rate(xxx/hr), 0-6h | ×× | ××× | ××× | ×× | ××× | ×× | ××× |
| Day 14 | Excretion Rate( $xxx/hr$ ), 0-4h | ××× | ××× | ××× | ××× | ××× | ××× | ××× |
| | Excretion Rate(xxx/hr), 4-8h | ××× | ××× | ××× | ××× | ××× | ××× | ××× |
| | Excretion Rate(xxx/hr), 8-12h | ××× | ××× | ××× | ××× | XXX | ××× | XXX |
| | Cumulative Excretion (xxx) | ××× | ××× | ××× | ××× | XXX | ××× | xxx |
| | Renal Clearance (mT./hr) | ××× | ××× | ××× | ××× | ××× | ××× | ××× |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas


Table 36. Summary Statistics of Estimated PK Urine Parameters for Ibudilast by Treatment STALICIA SA - Study No. STP1-C004
PK Population (N=xxxx)

Page x of y

Part 2 of 2: STP1- mg ibudilast

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Table 37. Summary Statistics of Estimated PK Urine Parameters for Bumetanide by Treatment STALICIA SA - Study No. STP1-C004
PK Population (N=xxx)

Page x of y

Part 1 of 2: STP1-Xmg ibudilast

| | | | | Day 14 | Day 1 | Visit |
|---|---|---|---|---|---|---|
| Renal Clearance (mL/hr) | Cumulative Excretion (xxx) | Excretion Rate(xxx/hr), 8-12h | Excretion Rate(xxx/hr), 4-8h | Excretion Rate( $xxx/hr$ ), 0-4h | Excretion Rate(xxx/hr), 0-6h | Parameter |
| ××× | ××× | ××× | ××× | ××× | ××× | B |
| ××× | ××× | ××× | ××× | ××× | ××× | Mean |
| xxx | ××× | ××× | ××× | ××× | ××× | Std Dev |
| ××× | ××× | ××× | ××× | ××× | ××× | CV% |
| xxx | ××× | ××× | ××× | ××× | ××× | Geometric<br>Mean |
| ××× | ××× | ××× | ××× | ××× | ××× | Lower<br>90% CI |
| ××× | ××× | ××× | ××× | ××× | ××× | Upper<br>90% CI |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas


Table 37. Summary Statistics of Estimated PK Urine Parameters for Bumetanide by Treatment STALICIA SA - Study No. STP1-C004
PK Population (N=xxx)

Page x of y

Part 2 of 2: STP1- mg ibudilast

| | | | | Day 14 | Day 1 | Visit |
|---|---|---|---|---|---|---|
| Renal Clearance (mL/hr) | Cumulative Excretion (xxx) | Excretion Rate(xxx/hr), 8-12h | Excretion Rate(xxx/hr), 4-8h | Excretion Rate(xxx/hr), 0-4h | Excretion Rate(xxx/hr), 0-6h | Parameter |
| ××× | ××× | ××× | ××× | ××× | ××× | n |
| XXX | ××× | ××× | ××× | ××× | ××× | Mean |
| ××× | ××× | ××× | ××× | ××× | XXX | Std Dev |
| XXX | ××× | ××× | ××× | ××× | ××× | CV% |
| XXX | ××× | ××× | ××× | XXX | XXX | Geometric<br>Mean |
| ××× | ××× | ××× | ××× | ××× | XXX | Lower<br>90% CI |
| ××× | ××× | ××× | ××× | ××× | ××× | Upper<br>90% CI |

Table 38. NIH-CTB Summary Statistics STALICLA SA - Study No. STP1-C004 Exploratory Population (N=xxx)

Page x of y

| ( | Overall | Placebo | | STP1-XXmg ibudilast | | | STP1-Xmg ibudilast | Treatment |
|---|---|---|---|---|---|---|---|---|
| 2222222 | ×××××××××××××××××××××××××××××××××××××× | ××××××××× | | ××××××××× | | | ××××××××× | Neurological<br>Function<br>Domain |
| XXXXXX | xxxxxx<br>xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Baseline | ××××× | Baseline | XXXXXX | ××××× | Baseline | Visit |
| RAW | RAW<br>CFB<br>RAW | RAW | RAW | RAW | CFB | RAW | RAW | Data<br>Type <sup>a</sup> |
| ××× | × | × ×<br>× × | ××× | ××× | ××× | ××× | ××× | n |
| XXX | × | × ×<br>× × | × | ××× | XXX | ××× | ××× | Mean |
| ××× | × | × ×<br>× × | ×× | ××× | ××× | ××× | ××× | Std<br>Dev |
| ××× | × ××<br>× ×× | × × | × | ××× | ××× | ××× | ××× | Median |
| ××× | × | × ×<br>× × | × | ××× | ××× | ××× | ×××× | Min |
| × × : | × ××<br>× ×× | × ×<br>× × | ××× | ××× | ××× | ××× | ××× | Max |

STATKING Clinical Services (month day, year) RAW = observed data recorded in database; CFB = change from baseline = (score at current visit) - (Baseline score).

Source Program: xxxxxxx.sas

Processing Speed Test Raw Score, Flanker Inhibitory Control and Attention Test Raw Score, Dimensional Change Card Sort Test Raw Score, Oral Reading Recognition Test Raw Score, Cognition Crystallized Composite Uncorrected Standard Score, Cognition Crystallized Composite Age-Corrected Standard Score, Cognition Crystallized National Percentile (Age Neurological Function Domain will include the following: Picture Vocabulary Test Raw Score, Pattern Comparison Adjusted), and Cognition Crystallized Composite Fully-Corrected T-score.

Table format will be repeated for KiTAP.


Table 40. OACIS-C Summary Statistics STALICLA SA - Study No. STP1-C004 Exploratory Population (N=xxx)

Page x of y

| 0 | ъ | ω | ω | н |
|---|---|---|---|---|
| Overall | Placebo | TP1-Xng | TP1-Xmg | Treatment |
| | | mg ibudilast | ng ibudilast | |
| *********** | *********** | *********** | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Question |
| × ×<br>× × | × × × × × | × ×<br>× × | × ×<br>× × | n |
| × ×<br>× × | × × × × × | × ×<br>× × | × ×<br>× × | Mean |
| × ×<br>× × | × ×<br>× × | × ×<br>× × | × ×<br>× × | Std Dev |
| × ×<br>× × | × ×<br>× × | × ×<br>× × | ×××<br>××× | Median |
| × ×<br>× × | × × × × × | × ×<br>× × | ××× | Min |
| × ×<br>× × | × × × × | × ×<br>× × | × × × × × | Max |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas


Page x of y

Table 41. Summary of Responses for OACIS-C Assessment by Question STALICIA SA - Study No. STP1-C004 Exploratory Population (N=xxx)

| Question General Level of Autism | Response Very Much Improved | ibu<br>(N | STP1 mg ibudilast (N=xxx) <sup>a</sup> xx (xxx) | STP1-<br>ibudi<br>(N=x | ibudilast (N=xxx) <sup>a</sup> xx (xxx) | Pla<br>(N=: | Placebo<br>(N=xxx) <sup>a</sup> |
|---|---|---|---|---|---|---|---|
| General Level of Autism | Very Much Improved<br>Much Improved<br>Minimally Improved | × × × | ( | × × × | ( ( ( X X X X X X X X X X X X X X X X X | × × × | * * * |
| | No Change | × > | (xxx) | × > | (×××) | × > | ( ( X X X ) |
| | Minimally Worse | × | (xxx) | × | (xxx) | × | |
| | Much Worse | ×× | (xxx) | × | (xxx) | × | (xxx) |
| | Very Much Worse | × | (xxx) | ×× | (xxx) | × | (xxx) |
| | Very Much Improved or Much | × | (xxx) | × | (xxx) | × | (xxx) |
| | Minimally Improved, No Change or Minimally Worse | × | (xxx) | × | (xxx) | xx (xxx) | _ |
| | Much Worse or Very Much Worse | × | (xxx) | × | (xxx) | × | (xxx) |
| Social Interaction Skills | Very Much Improved | ×× | (xxx) | ×× | (xxx) | × | (xxx) |
| | Much Improved | ×× | (xxx) | × | (xxx) | × | (xxx) |
| | Minimally Improved | × | (xxx) | × | (xxx) | × | (xxx) |
| | No Change | × | (xxx) | × | (xxx) | × | (xxx) |
| | Minimally Worse | × | (xxx) | × | (xxx) | ×× | (xxx) |
| | Much Worse | × | (xxx) | × | (xxx) | × | (xxx) |
| | Very Much Worse | × | (xxx) | × | (xxx) | × | (xxx) |
| | Very Much Improved or Much | × | (xxx) | × | (xxx) | × | (xxx) |
| | Improved Minimally Improved, No Change or Minimally Worse | × | (xxx) | × | (xxx) | × | (xxx) |
| | Much Worse or Very Much Worse | × | (xxx) | × | (xxx) | × | (xxx) |
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxxxxx | ×× | (xxx) | × | (xxx) | × | (xxx) |
| | XXXXXXXXXXXXX | ×× | () | | | 4 | |

The denominator for all proportions is the number of Exploratory population patients in the corresponding treatment group and overall. STATKING Clinical Services (month day, year)
Source Program: xxxxxxx.sas


| Exploratory Population (N=xxx) | STALICIA SA - Study No. STP1-C004 | Table 42. Summary of Responses for OACIS-S Assessment by Question | |
|---|---|---|---|
| | | | Page x of y |

| | ı | STP1-Xmg<br>ibudilast | STP1-\_ng ibudilast | Placebo | Overall |
|---|---|---|---|---|---|
| Question | Response | (N=xxx) a | (N=xxx) a | (N=xxx) a | (N=xxx) a |
| ××××××××××××××××××××××××××××××××××××××× | Normal | | | | |
| | Some symptom/ behavior | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| | Mild symptom/ behavior | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| | Moderate symptom/ behavior | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| | Marked symptom/ behavior | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| | Severe symptom/ behavior | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| | Among the Most Severe | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Normal | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx |
| | Some symptom/ behavior | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| | Mild symptom/ behavior | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx |
| | Moderate symptom/ behavior | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| | Marked symptom/ behavior | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| | Severe symptom/ behavior | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| | Among the Most Severe | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| xxxxxxxxxxxxxxxx | XXXXXXXXXXXX | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| | XXXXXXXXXXXX | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |

The denominator for all proportions is the number of Exploratory population patients in the corresponding treatment group and overall. STATKING Clinical Services (month day, year)
Source Program: xxxxxxx.sas


Table 43. ABC-C Summary Statistics STALICLA SA - Study No. STP1-C004 Exploratory Population (N=xxx)

Page x of y

| Overall | Placebo | | STP1ng<br>ibudilast | STP1-Xmg<br>ibudilast | Treatment |
|---|---|---|---|---|---|
| ×× | ×××××××××××××××××××××××××××××××××××××× | | × | XXXXXXXXXXXXXX | Subscale |
| xxxxxx<br>xxxxxx<br>xxxxxx | Baseline xxxxxx xxxxxx xxxxxx | ××××××××××××××××××××××××××××××××××××××× | xxxxxx Baseline xxxxxx | Baseline xxxxx xxxxx | Visit |
| RAW<br>CFB<br>RAW<br>CFB | RAW<br>RAW<br>CFB<br>RAW<br>CFB | RAW<br>CFB | CFB<br>RAW<br>RAW<br>CFB | RAW<br>RAW<br>CFB | Data<br>Type <sup>a</sup> |
| ×× ×××<br>×× ××× | ×× ×××<br>×× ××× | × ×<br>× × | × × × × × × × | × × × × × × | n |
| × | × | × ×<br>× × | × × × × × × × | × × × × × × × | Mean |
| × | ** *** | × × × × | × × × × × × × | × | Std Dev |
| × | * | ××× | × | × | Median |
| × | × | ××× | × × × × × × | XX | Min |
| × | × | × ×<br>× × | × | × | Max |

RAW = observed data recorded in database; CFB = change from baseline = (score at current visit) - (Baseline score). STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas


Table 44. SRS-2 Summary Statistics STALICLA SA - Study No. STP1-C004 Exploratory Population (N=xxx)

Page x of y

| | CV C | | | Placebo | | | ibudilast | STP1-Xng | | | \$<br>\$<br>\$<br>\$<br>\$ | STP1-Xmg | Treatment |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | > | | | XXXXXXXXXXXX | | | | ××××××××××××××××××××××××××××××××××××××× | | | | ****** | Subscale |
| ×××××<br>××××× | XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | × | Baseline<br>xxxxxx | XXXXXX | × | XXXXXX | Baseline | ××××× | ××××× | ×××××× | Baseline | Visit |
| RAW<br>CFB | RAW<br>CFB | CFB | CFB<br>RAW | RAW<br>RAW | CFB | CFB<br>RAW | RAW | RAW | RAW<br>CFB | CFB | RAW | RAW | Data<br>Type <sup>a</sup> |
| × ×<br>× × | × × × × | ××× | × ×<br>× × | × ×<br>× × | ××× | × × | ××× | ××× | × ×<br>× × | ××× | ××× | ××× | n |
| × ×<br>× × | × × × | ××× | × ×<br>× × | × ×<br>× × | ××× | × ×<br>× × | ××× | ××× | × ×<br>× × | ×× | ××× | ××× | Mean |
| × ×<br>× × | × × > | × | × ×<br>× × | ××× | ×× | × ×<br>× × | ××× | ××× | × ×<br>× × | ×× | ××× | ××× | Std Dev |
| × ×<br>× × | × × × × | XXX | X X<br>X X | × ×<br>× × | XXX | × ×× | ××× | ××× | × ×<br>× × | ××× | XXX | ××× | Median |
| × ×<br>× × | × × × × | ××× | X X<br>X X | × ×<br>× × | XXX | × ×<br>× × | ××× | ××× | × ×<br>× × | ×× | ××× | ××× | Min |
| × ×<br>× × | × × × × | XXX | X XX | × ×<br>× × | XXX | × × | ××× | ××× | × ×<br>× × | ××× | ××× | × | Max |

RAW = observed data recorded in database; CFB = change from baseline = (score at current visit) - (Baseline score). STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Table 45. Summary of Responses for CSHQ Assessment by Question STALICIA SA - Study No. STP1-C004 Exploratory Population (N=xxx)

Page x of y

| | | | STP1mg<br>ibudilast | STP1ng | Placebo | Overall |
|---|---|---|---|---|---|---|
| Visit | Question | Response | (N=XXX) a | (N=xxx) a | (N=xxx) a | (N=xxx) a |
| ××× | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Never | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| | | Rarely | xx (xxx) | xx (xxx) | xx (xxx) | ×× |
| | | Sometimes | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| | | Usually | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| | | Always | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| | ××××××××××××××××××××××××××××××××××××××× | Never | xx (xxx) | xx (xxx) | xx (xxx) | ×× |
| | | Rarely | xx (xxx) | xx (xxx) | xx (xxx) | XX ( |
| | | Sometimes | xx (xxx) | xx (xxx) | xx (xxx) | XX ( |
| | | Usually | xx (xxx) | xx (xxx) | xx (xxx) | ×× |
| | | Always | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ××××××××××××××××××××××××××××××××××××××× | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| | | | | () | ww (www) | ×× (××× |

The denominator for all proportions is the number of Exploratory population patients in the corresponding treatment group and overall. STATKING Clinical Services (month day, year)
Source Program: xxxxxxx.sas


Table 46. Lactate and Pyruvate Blood Level Summary Statistics STALICIA SA - Study No. STP1-C004 Exploratory Population (N=xxx)

Page x of y

| Treatment | Parameter (units) | Visit | Data<br>Type <sup>a</sup> | Þ | Mean | Std Dev | Min | Max | Median |
|---|---|---|---|---|---|---|---|---|---|
| STP1-Xmg | Lactate (xxx) | Baseline | RAW | ××× | ××× | ××× | ××× | ×<br>×<br>× | ××× |
| TENUTTASC | | ××××× | RAW | ××× | ××× | ××× | ××× | ××× | ××× |
| | | | CFB | ××× | ××× | ××× | ××× | ××× | ××× |
| | Pyruvate (xxx) | Baseline | RAW | ××× | ××× | ××× | ××× | ××× | ××× |
| | | XXXXXX | RAW | ××× | ××× | ××× | ××× | ××× | ××× |
| | | | CFB | ××× | ××× | ××× | ××× | ××× | ××× |
| | L:P Ratio (xxx) | Baseline | RAW | ××× | ××× | ××× | ××× | ××× | ××× |
| | | XXXXXX | RAW | ××× | ××× | ××× | ××× | ××× | ××× |
| | | | CFB | ××× | ××× | ××× | ××× | ××× | ××× |
| STP1-\mg | xxxxxxxxxx (xxx) | Baseline | RAW | ××× | ××× | ××× | ××× | ××× | ××× |
| 5 5 6 6 6 6 6 6 6 6 6 6 6 6 6 6 6 6 6 6 | | XXXXXX | RAW | ××× | ××× | ××× | XXX | ××× | ××× |
| | | | CFB | ××× | ××× | ××× | ××× | ××× | ××× |
| Placebo | xxxxxxxxxx (xxx) | Baseline | RAW | XXX | XXX | ××× | ××× | ××× | ××× |
| | | XXXXXX | RAW | ××× | ××× | ××× | ××× | ××× | ××× |
| | | | CFB | ××× | ××× | ××× | ××× | ××× | ××× |
| Overall | xxxxxxxxxx (xxx) | Baseline | RAW | XXX | XXX | XXX | XXX | ××× | ××× |
| | | XXXXXX | RAW | ××× | ××× | ××× | ××× | XXX | ××× |
| | | | CFB | XXX | XXX | ××× | ××× | XXX | XXX |
| bserved data; CFB = G Clinical Services | TB = change from baseline ices (DDMMMYYYY) | Ш | (results at current visit) - | visit) - | | (Baseline results). | | | |
| () HILLIAH () HILLIAH | | | | | | | | | |

Raw = observed data; CFB = change from STATKING Clinical Services (DDMMMYYYY) Source Program: xxxxxxxx.sas


Table 47. Summary of Responses for CGI-S Assessment by Visit STALICIA SA - Study No. STP1-C004 Exploratory Population (N=xxx)

Page x of y

| Visit | xxx Not Assessed | Normal, | Borderl | Mildly ill | Moderat | Markedly ill | Severely ill | Among t | patients | xxx Not Assessed | Normal, | Border | Mildly ill | Moderat | Markedly ill | Severely ill | Among t |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Response | | Normal, not at all ill | Borderline mentally ill | 111 | Moderately ill | ly ill | ly ill | Among the most extremely ill | C. C. | sessed | Normal, not at all ill | Borderline mentally ill | 111 | Moderately ill | ly ill | ly ill | Among the most extremely ill |
| $STP1-\underset{\text{ibudilast}}{\underbrace{\hspace{1cm}}} mg$ | ×× (×××) | xx (xxx) | (xxx) xx | xx (xxx) | xx (xxx) | (xxx) xx | xx (xxx) | xx (xxx) | | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| | | <u> </u> | <u> </u> | _ | _ | | | _ | | <u> </u> | _ | _ | _ | _ | | _ | |
| STP1-\text{ng ibudilast (N=xxx)} | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) | | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) | xx (xxx) |
| P1a | ×× | ×× | × | ×× | × | × | × | × | | × | × | ×× | × | ×× | ×× | × | × |
| Placebo<br>(N=xxx) <sup>a</sup> | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) |
| 0ve | × | × | × | ×× | × | ×× | ×× | ×× | | × | ×× | ×× | ×× | ×× | ×× | ×× | × |
| Overall | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) | (xxx) |

The denominator for all proportions is the number of Exploratory population patients in the corresponding treatment group and overall. STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas


Table 48. Summary of Responses for CGI-I Assessment by Visit STALICIA SA - Study No. STP1-C004 Exploratory Population (N=xxx)

Page x of y

| | | STP | STP1-Xmg | STP | STP1-X mg | Pl: | Placebo | Overall |
|---|---|---|---|---|---|---|---|---|
| Visit | Response | (N= | (N=xxx) a | (N | (N=XXX) a | (N= | (N=xxx) a | (N=xxx) a |
| ××× | Not assessed | × | (xxx) | × | (xxx) | × | (xxx) | × |
| | Very Much Improved | ×× | (xxx) | ×× | (xxx) | × | (xxx) | ×× |
| | Much Improved | × | (xxx) | ×× | (xxx) | × | (xxx) | ×× |
| | Minimally Improved | ×× | (xxx) | ×× | (xxx) | × | (xxx) | ×× |
| | No change from Baseline | × | (xxx) | ×× | (xxx) | × | (xxx) | ×× |
| | Minimally Worse | ×× | (xxx) | ×× | (xxx) | ×× | (xxx) | ×× |
| | Much Worse | ×× | (xxx) | ×× | (xxx) | ×× | (xxx) | ×× |
| | Very Much Worse | × | (xxx) | × | (xxx) | × | (xxx) | × |
| ××× | Not assessed | × | (xxx) | × | (xxx) | × | (xxx) | × |
| | Very Much Improved | ×× | (xxx) | ×× | (xxx) | ×× | (xxx) | ×× |
| | Much Improved | ×× | (xxx) | ×× | (xxx) | ×× | (xxx) | ×× |
| | Minimally Improved | ×× | (xxx) | ×× | (xxx) | ×× | (xxx) | ×× |
| | No change from Baseline | ×× | (xxx) | ×× | (xxx) | ×× | (xxx) | ×× |
| | Minimally Worse | × | (xxx) | ×× | (xxx) | × | (xxx) | ×× |
| | Much Worse | ×× | (xxx) | ×× | (xxx) | ×× | (xxx) | ×× |
| | Very Much Worse | ×× | (xxx) | ×× | (xxx) | ×× | (xxx) | ×× |

The denominator for all proportions is the number of Exploratory population patients in the corresponding treatment group and overall. STATKING Clinical Services (month day, year)
Source Program: xxxxxxx.sas

Table 49. Number and Proportion of Patients with Medical History Events STALICIA SA - Study No. STP1-C004
Safety Population (N=xxx) Page x of y

| Medical History Category <sup>a</sup> : | STP1-mg ibudilast (N=xxx)b | STP1————ng ibudilast (N=xxx) <sup>b</sup> | Placebo<br>(N=xxx) <sup>b</sup> | Overall (N=xxx) b |
|---|---|---|---|---|
| Total Number of Medical History Events | ××× | ××× | ××× | ××× |
| Patients with at Least One Medical History Event | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| System Organ Class 1 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 1 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 2 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| System Organ Class 2 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 1 | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) |
| Preferred Term 2 | xxx (xxx) | VVV (VVV) | xxx (xxx) | xxx (xxx) |

Source Program: xxxxxxx.sas


Medical history events coded with MedDRA Coding Dictionary Version XXX.

b The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall.

STATKING Clinical Services (month day, year)

Table 50. Number and Proportion of Patients Taking Concomitant Medications by ATC Level 4 and Preferred Page x of y

STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

| WHO Preferred Term 1 WHO Preferred Term 2 | ATC Level 4 Term | WHO Preferred Term 2 | WHO Preferred Term 1 | ATC Level 4 Term | Patients Taking at Least One Concomitant Medication | Total Number of Concomitant Medications | Concomitant Medication Category $^{\mathrm{a,b}}$ |
|---|---|---|---|---|---|---|---|
| xxx (xxx) | xxx (xxx) | | xxx (xxx) | xxx (xxx) | xxx (xxx) | ××× | $STP1-Mng$ ibudilast $(N=xxx)^{\circ}$ |
| xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | XXX | STP1-\_mg ibudilast (N=xxx)° |
| xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx | Placebo<br>(N=xxx)° |
| xxx (xxx) xxx | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx (xxx) | xxx | Overall<br>(N=xxx)° |

Source Program: xxxxxxx.sas

<sup>&</sup>lt;sup>a</sup> Concomitant medications coded with WHO Coding Dictionary xxxxxxxxxxxx.

<sup>b</sup> Concomitant medication category will include anatomical therapeutic chemical (ATC) level 4 term followed by preferred term.

<sup>c</sup> The denominator for all proportions is the number of Safety population patients in the corresponding treatment group and overall.

STARKING Clinical Services (month day, year)

Data Listing 1. Patient Disposition Data Listing STALICLA SA - Study No. STP1-C004

Page x of y

| ><br>><br>> | ×××× | XXXX | ×××× | Patient<br>No. |
|---|---|---|---|---|
| >>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>> | ×××××× | XXXXXX | ×××××× | Treatment |
| >>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>> | XXXXXX | XXXXXX | ×××××× | Date of<br>Informed<br>Consent |
| >>>>>> | XXXXXX | XXXXXX | XXXXXX | Date of<br>Randomization |
| >>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>> | XXXXXXXXX | XXXXXXXXXX | XXXXXXXXX | Disposition<br>Status |
| >>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>> | XXXXXXXX | XXXXXXXXX | XXXXXXXXX | Disposition<br>Date |
| >>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>> | XXXXXXXX | XXXXXXXXX | XXXXXXXX | Date of Last Visit/ Withdrawal Date |
| ********* | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXX | If Withdrawn, Reason for Discontinuation |
| *********** | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXX | If Discontinued from STP1, Reason for Discontinuation |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Data Listing 2. Demographics Data Listing STALICIA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| XXXX | xxxx | XXXX | xxxx | Patient<br>No. |
|--------|--------|--------|--------|-------------------------------|
| XXXXXX | XXXXXX | XXXXXX | ××××× | Treatment |
| XXXXXX | XXXXXX | XXXXXX | XXXXXX | Informed<br>Consent<br>Date |
| XXXXXX | XXXXXX | XXXXXX | XXXXXX | Date of<br>Birth |
| ××× | ××× | xxx | ××× | Age<br>(Years) |
| ××× | ××× | ××× | ××× | Height<br>(cm) |
| ××× | ××× | ××× | ××× | Weight (kg) |
| xxx | XXX | XXX | XXX | Two Years of |
| ××× | ××× | XXX | ××× | BMI |
| XXXXXX | xxxxxx | XXXXXX | xxxxxx | Gender |
| XXXXXX | XXXXXX | XXXXXX | xxxxxx | Ethnicity |
| XXXXXX | xxxxxx | XXXXXX | XXXXXX | Race |
| ×××××× | XXXXXX | XXXXXX | XXXXXX | SB5-<br>ABIQ<br>FSIQ<br>Score |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Data Listing 3. Adverse Events Data Listing STALICIA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

Part 1 of 2

| ×<br>×<br>×<br>×<br>×<br>×<br>× | ××××××× | Patient<br>No. |
|---|---|---|
| ×<br>×<br>×<br>×<br>× | × | Treatment |
| ×<br>×<br>×<br>×<br>× | ×××××× | Treatment<br>Start Date |
| ******* | ********/ | AE Start<br>Date/<br>AE End<br>Date |
| ************************************** | ************************************** | MedDRA System Organ Classa/ MedDRA Preferred Term/ CRF Verbatim Term |
| ×<br>×<br>×<br>×<br>×<br>× | ××××××× | Severity |
| ××××××××××××××××××××××××××××××××××××××× | ××××××× | AE of<br>Special<br>Interest? |
| ×<br>×<br>×<br>×<br>×<br>× | ××××××× | Relationship<br>to Study<br>Drug |
| **/ | **/ | Serious? (Y/N)/ Reason Serious? |

Adverse events coded with MedDRA Coding Dictionary Version xxx. STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas


Data Listing 3. Adverse Events Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

Part 2 of 2

| xxxxxxxx | ××××××××××××××××××××××××××××××××××××××× | Patient<br>No. |
|---|---|---|
| ××××× | ×××××× | Treatment |
| ×××××× | ××<br>××<br>××<br>×× | Treatment<br>Start Date |
| ******* | ******** | AE Start Date/ AE End Date |
| ************************************** | ************************************** | MedDRA System Organ Classa/ MedDRA Preferred Term/ CRF Verbatim Term |
| ×××× | ×××× | Action<br>Taken |
| ××××××× | ×<br>×<br>×<br>×<br>×<br>× | Outcome |
| xxx | ××× | Led to Study Treatment Discontinuation (Y/N)? |

Adverse events coded with MedDRA Coding Dictionary Version xxx. STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas


Data Listing 4. Vital Signs Data Listing STALICIA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| ××××× | Patient<br>No. |
|--------------|----------------------------------|
| ××××<br>×××× | Treatment |
| XXXXXX | Treatment<br>Start Date |
| ***** | Visit |
| ***** | Visit<br>Date |
| ×××××× | Time |
| ***** | Patient<br>Position <sup>a</sup> |
| ×××××× (×××) | Parameter<br>(Units) |
| ***** | Result |

Patient position will distinguish between supine blood pressure and heart rate and standing blood pressure and heart rate. STATKING Clinical Services (month day, year)
Source Program: xxxxxxx.sas


Data Listing 5. Baseline ECG Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

Part 1 of 2

| No. | 2000 | | |
|-----------|--------|------|------|
| Treatment | 000000 | | |
| of ECG | 200000 | | |
| Time | 2000 | XXXX | XXXX |
| HR | 200 | ××× | XXX |
| PQ | 200 | XXX | ××× |
| Duration | 2000 | ×××× | XXXX |
| Interval | 2000 | ×××× | XXXX |
| RR | 200 | ×× | ×× |
| QTCF | 2000 | xxxx | XXXX |

The Day 1 prior to treatment (i.e., pre-dose) time point serves as baseline. STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Data Listing 5. Baseline ECG Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

Part 2 of 2

| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|------------------------------|----------------------------------------------|
| XXXX XXXX | XXXX XXXX XXXX XXXXX XXXXX |
| | XXXXXXX<br>XXXXXXXX<br>XXXXXXXX |
| ××××××<br>×××××××<br>××××××× | |
| | ××××××<br>×××××××<br>××××××××××××××××××××××× |

The Day 1 prior to treatment (i.e., pre-dose) time point serves as baseline. STATKING Clinical Services (month day, year)
Source Program: xxxxxxxx.sas

Data Listing 6. ECG Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

Part 1 of 2

| | | | | ı | | |
|-------|--------|-------|--------|-------------|-----------|-----------------|
| | ×××× | | ×××× | No. | Patient | |
| | xxxxxx | | XXXXXX | Treatment | | |
| | ××××× | | ××××× | Visit | | |
| | ×××××× | | ×××××× | ECG | Date of | |
| XXXXX | xxxxx | XXXXX | XXXXX | Post-Dose | Pre-Dose/ | |
| ×××× | ×××× | ×××× | XXXX | Time | | |
| ×××× | ×××× | XXXX | ×××× | HR | | |
| ×××× | ×××× | XXXX | ×××× | PΩ | | |
| ×××× | ×××× | ×××× | XXXX | PQ Duration | QRS | ECG Parametersa |
| ×××× | ×××× | xxxx | ×××× | Interval | ΩĦ | metersa |
| × | × | × | × | RR | | |
| ×××× | ×××× | ×××× | ×××× | QTCF | | |

ECG parameters and results for T Wave, U Wave and ECG Interpretation displayed at Baseline (i.e., Day 1 pre-dose time point) are the average and combined overall results.

STATKING Clinical Services (month day, year)

Source Program: xxxxxxxx.sas


Data Listing 6. ECG Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

Part 2 of 2

Patient ×××× XXXX Treatment ××××× XXXXXX Visit XXXXX XXXXX Date of ECG ×××××× XXXXXXX Pre-Dose/ Post-Dose × Time × × × × × × X X X X X X T Wave × U Wave × ECG Resultsa Interpretation × ECG Significant (Y/N)? Abnormal, Clinically ××××××× ××××××× ××××××× xxxxxxx Ιf XXXXXXXXXX XXXXXXXXXX XXXXXXXXXX XXXXXXXXXX Description

Source Program: xxxxxxx.sas

<sup>&</sup>lt;sup>a</sup> ECG parameters and results for T Wave, U Wave, and ECG Interpretation displayed at Baseline (i.e., Day 1 pre-dose time point) are the average and combined overall results.

STATKING Clinical Services (month day, year)

Data Listing 7. Blood Chemistry Laboratory Results Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| ×××× | ×××× | Patient<br>No. |
|---|---|---|
| XXXXXX | xxxxxx | Treatment |
| ××××× | ×××× | Visit |
| ××××× | ××××× | Date of<br>Visit |
| xxxxxxxxx (xxx) | xxxxxxxxx (xxx) | Parameter (units) |
| XXX | ××× | Result |
| ××× | × | Norma |
| ××× | ××× | Normal Range<br>Low High |
| ×××× | xxxxx | Normal/High/Low <sup>a</sup> |
| ××××××××× | ×××××××× | Normal/Abnormal CS/<br>Abnormal NCS <sup>b</sup> |

normal range. Indicates whether the results of the parameter indicated were within the normal range, lower than the normal range, or higher than the

b Indicates whether the results of the parameter indicated were Normal, Abnormal Clinically Significant (CS), and Abnormal Not Clinically Significant (NCS).

STATKING Clinical Services (month day, year)

Source Program: xxxxxxxx.sas

Data Listing 8. Serology Laboratory Results Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| | | ı |
|-----------|-----------|------------------|
| ×××× | ×××× | Patient<br>No. |
| ×××××× | XXXXXX | Treatment |
| xxxxxx | xxxxxx | Visit |
| ××××× | XXXXXX | Date of<br>Visit |
| xxxxxxxxx | XXXXXXXXX | Parameter ( |
| (xxx) | (xxx) | (units) |
| XXX | ××× | Result |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Data Listing 9. Hematology Laboratory Results Data Listing STALICIA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| | XXXX XXXXXX XXXXXXX XXXXXXXXXXXXXXXXXX | Patient No. Treatment Visit Visit Parameter (units) Result Low Hig |
|---|---|---|
| xxxxxxxxx (xxx) xxx | | |
| ××× | ××× | Tow |
| ××× | ××× | High |
| ××××× | ×××× | Normal/High/Low <sup>a</sup> |

Indicates whether the results of the parameter indicated were within the normal range, lower than the normal range, or higher than the normal range.

STATKING Clinical Services (month day, year)

Source Program: xxxxxxx.sas

Listing format repeats for Coagulation and Urinalysis.

Data Listing 12. Hearing Assessment Data Listing STALICLA SA - Study No. STP1-C004

Page x of y

| Patient No. Treatment Visit Visit Since last visit? | Safety Population (N=xxx) |
|---|---|
|---|---|

XXXX XXXX

XXXXXX XXXXXX

XXXXXX XXXXXX

XXXXXX XXXXXX

××× ×××

XXXXXXXXXX XXXXXXXXXX

STATKING Clinical Services (month day, year)
Source Program: xxxxxxxx.sas

Data Listing 13. Pharmacokinetic Blood Sample Data Listing STALICLA SA - Study No. STP1-C004 PK Population (N=xxx)

Page x of y

| | ×××× | | ×××× | Patient<br>No. |
|---------|---------|---------|---------|----------------------------------|
| | ××××× | | ×××××× | Treatment |
| | ×××× | | ×××× | Visit |
| | ***** | | ***** | Dose<br>Date/<br>Time |
| | ××× | | ××× | Blood Draw<br>Completed<br>(Y/N) |
| | ××××××× | | ××××××× | Reason<br>Not<br>Completed |
| XXXXXXX | XXXXXXX | xxxxxxx | ××××××× | Time<br>Point |
| ×××× | ×××× | XXXX | ×××× | Time of<br>Blood<br>Sample |
| ×××× | ×××× | XXXX | ×××× | Time of Plasma Extraction |
| ×××× | ×××× | ×××× | ×××× | Time of<br>Aliquot<br>Freezing |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Data Listing 14. Pharmacokinetic Urine Sample Data Listing STALICLA SA - Study No. STP1-C004 PK Population (N=xxx)

Page x of y

| | XXXX | | ×××× | Patient<br>No. |
|---------|----------|----------|----------|----------------------------------|
| | ××××× | | ××××× | Treatment |
| | ×××× | | ×××× | Visit |
| | ×××××/ | | *****/ | Dose<br>Date/<br>Time |
| | ××× | | ××× | Urine Collection Completed (Y/N) |
| | ×××××××× | | ×××××××× | Reason<br>Not<br>completed |
| ××××××× | XXXXXXX | XXXXXXXX | ××××××× | Time<br>Point |
| xxxx | ×××× | ×××× | ×××× | Time of<br>Urine<br>Sample |
| ×××× | ×××× | ×××× | ×××× | Urine<br>Volume<br>(mL) |
| ×××× | ×××× | ×××× | ×××× | Time of<br>Aliquot<br>Freezing |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Data Listing 15. Plasma Concentrations Data Listing STALICIA SA - Study No. STP1-C004 PK Population (N=xxx)

Page x of y

| | ×××× | | XXXX | Patient<br>No. |
|---|---|---|---|---|
| | ××××× | | XXXXXX | Treatment |
| | ×××× | | ×××× | Visit |
| XXXXXXX | XXXXXXX | XXXXXXXX | XXXXXXXX | Time<br>Point |
| ×××× | ×××× | ×××× | ×××× | Sample Collected(Y/N)? |
| xxxx/xxxx | xxxx/xxxx | xxxx/xxxx | xxxx/xxxx | Sample Collected(Y/N)? Sample Date/ Time |
| xxxxxxx (xxx) | xxxxxxx (xxx) | xxxxxxx (xxx) | xxxxxxx (xxx) | Ibudilast Plasma Concentration (units) |
| xxxxxxx (xxx) | xxxxxxx (xxx) | xxxxxxx (xxx) | xxxxxxx (xxx) | Bumetanide Plasma<br>Concentration<br>(units) |

Data Listing 16. Urine Concentrations Data Listing STALICLA SA - Study No. STP1-C004 PK Population (N=xxx)

Page x of y

| | ×××× | | XXXX | Patient<br>No. |
|---|---|---|---|---|
| | xxxxxx | | XXXXXX | Treatment |
| | xxxx | | ××× | Visit |
| XXXXXXX | ××××××× | XXXXXXX | XXXXXXXX | Time<br>Interval |
| ×××× | ×××× | ×××× | ×××× | Sample Collected(Y/N)? |
| xxxx/xxxx | xxxx/xxxx | xxxx/xxxx | xxxx/xxxx | Sample<br>Date/Time |
| xxxxxxx (xxx) | xxxxxxx (xxx) | xxxxxxx (xxx) | xxxxxxx (xxx) | Ibudilast Urine Concentration (units) |
| xxxxxxx (xxx) | xxxxxxx (xxx) | xxxxxxx (xxx) | xxxxxxx (xxx) | Bumetanide Urine Concentration (units) |

Data Listing 17. Plasma Pharmacokinetics Parameters Data Listing STALICLA SA - Study No. STP1-C004 PK Population (N=xxx)

Page x of y

| Patient<br>No. | Treatment | Visit | Drug | Parameter (units) | Value |
|----------------|-----------|-------|-------|--------------------|-------|
| ××××× | xxxx | ××××× | xxxxx | xxxxxxxxxxx (xxx) | ××× |
| | | | | xxxxxxxxxx (xxx) | ××× |
| | | | | xxxxxxxxxx (xxx) | ××× |
| | | | | xxxxxxxxxxx (xxx) | XXX |
| XXXXX | XXXX | XXXXX | XXXXX | xxxxxxxxxxx (xxx) | ××× |
| | | | | xxxxxxxxxxx (xxx) | xxx |
| | | | | xxxxxxxxxxx (xxx) | ××× |
| | | | | xxxxxxxxxxxx (xxx) | ××× |
| XXXXX | ×××× | XXXXX | ××××× | xxxxxxxxxxxx (xxx) | ××× |
| | | | | xxxxxxxxxxx (xxx) | ××× |
| | | | | xxxxxxxxxxx (xxx) | xxx |
| | | | | xxxxxxxxxxx (xxx) | ××× |
| XXXXX | XXXX | XXXXX | XXXXX | xxxxxxxxxxx (xxx) | ××× |
| | | | | xxxxxxxxxxx (xxx) | ××× |
| | | | | xxxxxxxxxxx (xxx) | ××× |
| | | | | XXXXXXXXXXX (XXX) | ××× |

STATKING Clinical Services (month day, year) Source Program: xxxxxx.sas

Data Listin 18 11717 D' ioki n

| | | þ |
|---|---|---|
| | | Listing |
| | ß | _ |
| PK | TALICLA | Urine |
| PK Population | SA - Study | Pharmacokine |
| (N=xxx) | STALICLA SA - Study No. STP1-C004 | a Listing 18. Urine Pharmacokinetics Parameters Data Listing |

Page x of y

| Patient<br>No. | Treatment | Visit | Drug | Parameter (units) | Value |
|---|---|---|---|---|---|
| ×××× | ×××× | ××××× | XXXXX | xxxxxxxxxxx (xxx) | ××× |
| | | | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | ××× |
| | | | | xxxxxxxxxxx (xxx) | ××× |
| | | | | xxxxxxxxxxx (xxx) | ××× |
| XXXXX | XXXX | XXXXX | XXXXX | xxxxxxxxxxx (xxx) | ××× |
| | | | | xxxxxxxxxxx (xxx) | XXX |
| | | | | xxxxxxxxxxx (xxx) | ××× |
| | | | | xxxxxxxxxxx (xxx) | ××× |
| XXXXX | ×××× | XXXXX | ×××× | xxxxxxxxxxx (xxx) | ××× |
| | | | | xxxxxxxxxxx (xxx) | ××× |
| | | | | xxxxxxxxxxx (xxx) | xxx |
| | | | | xxxxxxxxxxx (xxx) | ××× |
| XXXXX | XXXX | XXXXX | XXXXX | xxxxxxxxxxx (xxx) | xxx |
| | | | | xxxxxxxxxxx (xxx) | xxx |
| | | | | xxxxxxxxxxx (xxx) | ××× |
| | | | | XXXXXXXXXXX (XXX) | ××× |

STATKING Clinical Services (month day, year) Source Program: xxxxxx.sas

Page x of y

| Safety Population (N=xxx) | STALICLA SA - Study No. STP1-C004 | Data Listing 19. C-SSRS Data Listing |
|---|---|---|

| | × | | ×××× | Patient No. |
|---|---|---|---|---|
| | ×<br>×<br>×<br>×<br>× | | ×××××× | Treatment |
| ×××× | ××× | ××× | ×××× | Visit |
| ××× | ××× | ××× | ×××× | Date |
| ************************************** | ************************************** | ************************************** | ************************************** | Question |
| × × ×<br>× × ×<br>× × × | × × ×<br>× × ×<br>× × × | × × ×<br>× × ×<br>× × × | × × ×<br>× × ×<br>× × × | Response |

STATKING Clinical Services (month day, year)
Source Program: xxxxxxxx.sas

Da:

Page x of y

| STALICIA SA - Study No. STP1-C004 Safety Population (N=xxx) |
|-------------------------------------------------------------|
|-------------------------------------------------------------|

| | ×××× | | ×××× | Patient No. |
|---|---|---|---|---|
| | ××××××××××××××××××××××××××××××××××××××× | | ××××× | Treatment |
| ××× | ××× | ××× | ×××× | Visit |
| ×××× | ×××× | ××× | ×××× | Date |
| ************************************** | ************************************** | ************************************** | ************************************** | Question |
| × × ×<br>× × ×<br>× × × | × | × × ×<br>× × ×<br>× × × | × × ×<br>× × ×<br>× × × | Response |

STATKING Clinical Services (month day, year)
Source Program: xxxxxxxx.sas


Data Listing 21. STALICLA SA -Safety Pop

| Population | - Study 1 | 21. OACIS- |
|------------|---------------|-----------------|
| n (N=xxx) | No. STP1-C004 | -S Data Listing |

Page x of y

| | | | | | | | | | XXXX | | | | | | | | | | ×××× | Patient No. |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | XXXXXX | | | | | | | | | | XXXXXX | Treatment |
| | | | | | | | | | ×××× | | | | | | | | | | XXXX | Visit |
| | | | | | | | | | ×××× | | | | | | | | | | XXXX | Date |
| XXXXXXXXXXXX | XXXXXXXXXXXXX | ××××××××××××××××××××××××××××××××××××××× | XXXXXXXXXXXXX | XXXXXXXXXXXX | XXXXXXXXXXXX | XXXXXXXXXXXXX | XXXXXXXXXXXXX | XXXXXXXXXXXXX | XXXXXXXXXXXXX | XXXXXXXXXXXX | XXXXXXXXXXXXX | XXXXXXXXXXXX | XXXXXXXXXXXXX | XXXXXXXXXXXX | XXXXXXXXXXXXX | XXXXXXXXXXXXX | XXXXXXXXXXXX | XXXXXXXXXXXXX | XXXXXXXXXXXX | Question |
| XXXX | XXXX | ×××× | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | xxxx | xxxx | XXXX | XXXX | XXXX | XXXX | XXXX | ×××× | XXXX | XXXX | XXXX | Response |

STATKING Clinical Services (month day, year)
Source Program: xxxxxxxx.sas

Data ST

Page x of y

| Safety Population | TALICLA SA - Study No. | a Listing 22. OACIS-C |
|-------------------|------------------------|-----------------------|
| (N=xxx) | STP1 | Data Listing |

| xxxxxx xxxx xxxx Social Interaction Skills Aberrant/Abnormal Behavior Repetitive and Ritual Behaviors Verbal Communication Skills | | Hyperactivity and Inattention Anxiety and Fears Anxiety and Fears Sensory Sensitivities Restricted and Narrow Interests General Level of Autism Social Interaction Skills Aberrant/Abnormal Behavior Repetitive and Ritual Behavior Verbal Communication Skills Nonverbal Communication Skills Hyperactivity and Inattention Anxiety and Fears | ×××× | × | ×<br>×<br>×<br>× | ×××× |
|---|---|---|---|---|---|---|
| xxxxxx xxxx xxxx General Level of Addism | : | Social Interaction Skills Aberrant/Abnormal Behavior Repetitive and Ritual Behaviors Verbal Communication Skills Verbal Communication Skills | | | | |
| | ×××× | General Level of Autism | XXXX | XXXX | ×××××× | ×××× |

STATKING Clinical Services (month day, year)
Source Program: xxxxxxx.sas

Page x of y

Treatment XXXXXX XXXXXX Visit ××××× ××××× ××××× ××××× Date Data Listing 23. SRS-2 Data Listing STALICIA SA - Study No. STP1-C004 Safety Population (N=xxx) ××××× ××××× Time Global Score × Social Awareness × Social Cognition XXXX XXXX × × × × × × Social Communication × Social Motivation × × × × × × XXXX XXXX Mannerisms × × × × × × ×××× XXXX

Patient No.

XXXX

XXXX

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Data Listing 24. SB5 ABIQ Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| xxxx | XXXX | Patient No. |
|--------|--------|--------------------------------------------|
| ×××××× | XXXXXX | Treatment |
| ×××× | ×××× | Date |
| xxxx | ×××× | Abbreviated IQ Test |
| xxxx | XXXX | IQ Test Performed with Last 2 years? (Y/N) |
| ×××× | ×××× | FSIQ Score |

STATKING Clinical Services (month day, year)
Source Program: xxxxxxxx.sas

Data Listing 25. NIH-CTB Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| | ×××× | | | | ×××× | Patient No. |
|---|---|---|---|---|---|---|
| | xxxxxx | | | | xxxxxx | Treatment |
| | ×××× | | ×××× | | ×××× | Visit |
| | ×××× | | ×××× | | ××× | Date |
| xxxxxxxxxxx | xxxxxxxxxxx | xxxxxxxxxxx | xxxxxxxxxxx | xxxxxxxxxxx | xxxxxxxxxxxx | Neurological<br>Function Domain |
| ×××× | ×××× | ×××× | ×××× | ×××× | xxxx | Score |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Processing Speed Test Raw Score, Flanker Inhibitory Control and Attention Test Raw Score, Dimensional Change Card Sort Test Raw Score, Oral Reading Recognition Test Raw Score, Cognition Crystallized Composite Uncorrected Standard Score, Cognition Crystallized Composite Age-Corrected Standard Score, Cognition Crystallized National Percentile (Age Neurological Function Domain will include the following: Picture Vocabulary Test Raw Score, Pattern Comparison Adjusted), and Cognition Crystallized Composite Fully-Corrected T-score.

Listing format repeats for KiTAP.

STATKING Clinical Services
Version 1.1


Data Listing 27. ABC-C Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| | ×××× | | XXXX | Patient No. |
|------|--------|------|--------|--------------------------------------|
| | XXXXXX | | XXXXXX | Treatment |
| ×××× | ×××× | ×××× | xxxx | Visit |
| ××× | ×××× | ×××× | xxxx | Date |
| ×××× | ×××× | ×××× | XXXX | Time |
| ×××× | ×××× | ×××× | XXXX | Irritability |
| ×××× | XXXX | XXXX | XXXX | Social<br>Withdrawal |
| ×××× | XXXX | XXXX | XXXX | Subscales<br>Stereotypic<br>Behavior |
| ×××× | ×××× | ×××× | ×××× | Hyperactive/<br>Noncompliance |
| ×××× | ×××× | ×××× | ×××× | Inappropriate<br>Speech |


Da S1

Page x of y

| | | ×××× | Patient No. |
|---|---|---|---|
| | | ××××× | Treatment |
| ×××× | ×××× | ×××× | Visit |
| XXXX | ×××× | ××× | Date |
| ××××××××××××××××××××××××××××××××××××××× | ××××××××××××××××××××××××××××××××××××××× | ****** | Category |
| ************************************** | ************************************** | ************************************** | Question |
| × × ×<br>× × ×<br>× × × | × × ×<br>× × ×<br>× × × | X | Response |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |


STALICLA SA February 17, 2022

Data Listing 29. Lactate-Pyruvate Data Listing STALICIA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| | | ъ | |
|----------|---------|-------------|----------|
| ×××× | ×××× | Patient No. | |
| ×××××× | ××××× | Treatment | |
| XXXXXXXX | ××××××× | Visit | |
| XXXXXXXX | ××××××× | Visit | Date of |
| XXXXXXXX | ××××××× | (units) | Taccace |
| XXXXXXX | ×××××× | (units) | FYLUVALE |
| XXXXXXX | ×××××× | Ratio | L., |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas
Data Listing 30. CGI-S/CGI-I Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| | XXXX | Patient No. Treatment |
|----------|----------|-----------------------|
| | XXXXXX | |
| XXXXXXX | XXXXXXXX | Visit |
| XXXXXXXX | XXXXXXXX | Visit Date of Visit |
| XXXXXXXX | XXXXXXXX | Severity of Illness |
| XXXXXXXX | | Global Improvement |

STATKING Clinical Services (month day, year) Source Program: xxxxxxxx.sas


Data Listing 31. Medical History Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| ×××××× | ××××× | Patient<br>No. |
|---|---|---|
| XXXXXXX | ×<br>×<br>×<br>×<br>× | Treatment |
| ************************************** | ************************************** | MedDRA System Organ Classa/<br>MedDRA Preferred Term/<br>CRF Verbatim Term |
| ××××××××××××××××××××××××××××××××××××××× | ×<br>×<br>×<br>×<br>× | Start Date |
| ××××××××××××××××××××××××××××××××××××××× | ××××××××××××××××××××××××××××××××××××××× | End Date |
| ×<br>× | ×<br>× | Ongoing? |

Medical history terms coded with MedDRA Coding Dictionary Version xxx. STATKING Clinical Services (month day, year)
Source Program: xxxxxxx.sas


Data Listing 32. Concomitant Medications Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| ××× | × | Pat |
|---|---|---|
| XXXXXX | xxxxxxx | Patient<br>No. |
| ××××× | xxxxx | Treatment |
| ************************************** | ************************************** | WHO Preferred Term*/ Verbatim Drug Name/ Indication/ ATC Level 4 Term |
| (xxx) | (xxx) | Dose<br>(units) |
| ×××××× | xxxxxxx | Frequency |
| XXXXXX | ××××××××××××××××××××××××××××××××××××××× | Start |
| ×××××× | ××××××××××××××××××××××××××××××××××××××× | Stop |
| ×<br>×<br>× | ×<br>×<br>×<br>× | Route |
| ×××××× | xxxxxx | Ongoin Ondication (Y/N) |
| ×××× | ×××× | Ongoing? |

Concomitant medication coded with WHO Coding Dictionary xxxxxxxxxx STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas


Data Listing 33. Physical Exam Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| Patient<br>No. | Treatment | Visit | Date | Body System | Result | If Abnormal, Clinically Significant (Y/N)? | |
|---|---|---|---|---|---|---|---|
| XXXX | XXXXXX | XXXXXXX | ×××××× | ××××××××××× | ×××××××× | ××××××× | |
| | | | | XXXXXXXXXXX | XXXXXXXX | XXXXXXX | |
| | | | | XXXXXXXXXXX | XXXXXXXX | xxxxxxx | ^ |
| | | XXXXXXX | XXXXXXX | XXXXXXXXXXX | XXXXXXXX | XXXXXXX | × |
| | | | | XXXXXXXXXXX | XXXXXXXX | XXXXXXX | × |
| | | | | XXXXXXXXXXX | XXXXXXXX | XXXXXXX | × |
| | | | | XXXXXXXXXXX | XXXXXXXX | xxxxxxx | × |
| | | | | XXXXXXXXXXX | XXXXXXXX | XXXXXXX | × |
| | | | | XXXXXXXXXXX | XXXXXXXX | XXXXXXX | × |
| | | | | XXXXXXXXXXX | ××××××× | XXXXXXX | ^ |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Data Listing 34. Study Drug Administration Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| ×××× | ×××× | Patient<br>No. |
|-------------|------------|--------------------------------------------|
| ××××× | ××××× | Treatment |
| XXXX | ×××× | Visit |
| ××× | ×××<br>××× | Morning Dose Administered (Y/N)? |
| *********** | ********** | Reason Morning<br>Dose Not<br>Administered |
| ****** | ****** | Date Morning Dose<br>Administered |
| ****** | XXXXXXX | Time Morning Dose<br>Administered |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas


Data Listing 35. Drug Accountability Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| ×××× | ×××× | Patient<br>No. |
|---|---|---|
| ××××× | ××××× | Treatment |
| × | × | Visit |
| ***** | ×××××××××××××××××××××××××××××××××××××× | Study Drug<br>Dispensed<br>Kit Number |
| ****** | ××××××<br>××××××××××××××××××××××××××××××× | Date Study<br>Drug<br>Dispensed |
| ***** | ×××××<br>×××××× | Number of<br>Pills<br>Dispensed |
| ***** | ××××××<br>××××××× | Study Drug<br>Returned<br>Kit Number |
| ***** | ×××××<br>×××××× | Date Study<br>Drug<br>Returned |
| ***** | ×××××××××××××××××××××××××××××××××××××× | Number of<br>Pills<br>Returned |
| × × × × | × ×<br>× × | Did Patient Take Study Medication as Directed (Y/N)? |
| ************************************** | XXXXXXX | Did Patient Take Study Medication as Directed If No, Please (Y/N)? Specify |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Data Listing 36. Urine Pregnancy Test Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| | | | | Pat: | | |
|---|---|---|---|---|---|---|
| | XXXX | | XXXX | Patient No. | | |
| | XXXXXX | | XXXXXX | Treatment | | |
| XXXXXX | XXXXXX | XXXXXX | XXXXXX | Visit | | |
| ××××× | ×××××× | ××××× | XXXXXX | Required? (Y/N) | Pregnancy Test | |
| XXXXXX | ×××××× | XXXXXX | XXXXXX | Performed? (Y/N) | Pregnancy Test | |
| XXXXXXXXX | XXXXXXXXX | XXXXXXXXX | XXXXXXXXX | Not Performed | Pregnancy Test | Reason |
| XXXXXXXXX | XXXXXXXXX | XXXXXXXXX | XXXXXXXXX | Test | of Pregnancy | Date and Time |
| XXXXXX | XXXXXX | XXXXXX | XXXXXX | Test | Pregnancy | Result of |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Data Listing 37. Protocol Deviations Data Listing STALICLA SA - Study No. STP1-C004 Safety Population (N=xxx)

Page x of y

| × | xxxx | Patient<br>No. |
|---|---|---|
| ****** | XXXXXX | Treatment |
| ***** | XXXXXX | Date of<br>Deviation |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Deviation Description |
| × | XXXXXXXX | Deviation Major or<br>Minor |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas


Data Listing 38. Patients Excluded from Safety Population Data Listing STALICIA SA - Study No. STP1-C004
All Patients (N=xxx)

Page x of y

| XXXX | XXXX | XXXX | XXXX | Patient No. |
|---|---|---|---|---|
| XXXXXX | XXXXXX | ×××××× | XXXXXX | Treatment |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ***** | Reason for Exclusion |

STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Data listing will be repeated for the PK and Exploratory populations.


Figure 1. Orthostatic Vital Signs - Spaghetti Plot of Systolic Blood Pressure by Patient, Time and STALICLA SA - Study No. STP1-C004 Treatment

Safety Population (N=xxx)

Page x of y



STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Note: the axis values and labels will vary depending on the figure generated and the data in the database. Patient ID's will be displayed as in the study database. Figure format will be repeated for Orthostatic Vital Signs - Diastolic Blood Pressure (Figure 2), Orthostatic Vital Signs - Heart Rate (Figure 3), ECG Parameters - Heart Rate (Figure 4), and ECG Parameters - QTCF (Figure 5).


Figure 6. Blood Chemistry - Spaghetti Plot of Sodium by Patient, Time and Treatment STALICLA SA - Study No. STP1-C004
Safety Population (N=xxx)

Page x of y



STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Figure format will be repeated for Figure format will be repeated for Blood Chemistry - Chloride (Figure 7), Blood Chemistry - Calcium (Figure 8), Blood Chemistry - Magnesium (Figure 9), Blood Chemistry - Phosphate (Figure 10), Blood Chemistry - Potassium (Figure 11), Hematology - Platelet Count (Figure 12), and Biomarker - L:P Ratio (Figure 13). Note: the axis values and labels will vary depending on the figure generated and the data in the database. Patient ID's will be displayed as in the study database.





STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

Figure format will be repeated for the 10mg ibudilast treatment group for ibudilast concentration levels, for the mg mg ibudilast treatment groups for bumetanide concentration levels. These figures will be repeated in the semi-logarithmic scale for each combination of treatment group and study drug concentration level.

Note: the axis values and labels in the figure may vary. Patient ID's will be displayed as in the study database.





STATKING Clinical Services (month day, year) Source Program: xxxxxxx.sas

logarithmic scale for each combination of treatment group and study drug concentration level.

the axis values and labels in the figure may vary. Figure format will be repeated for the 10mg ibudilast treatment group for ibudilast concentration levels, for the 5mg and 10mg ibudilast treatment groups for bumetanide concentration levels. These figures will be repeated in the semi-Note:


# **DocuSign**

**Certificate Of Completion** 

Envelope Id: 8C4D2141974A4A22BCBAF80DF8665E44

Subject: 20220218\_STALICLA\_STP1-C004\_Statistical Analysis Plan\_V1.1\_FINAL.docx Please DocuSign

Source Envelope:

Document Pages: 121
Certificate Pages: 5
AutoNav: Enabled

Envelopeld Stamping: Disabled

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Signatures: 4

Initials: 0

Envelope Originator: Mark Tetrick 759 Wessel Dr.

Fairfield, OH 45014

Status: Completed

mtetrick@statkingclinical.com IP Address: 216.196.246.214

**Record Tracking** 

Status: Original

February 18, 2022 | 08:53

Holder: Mark Tetrick

mtetrick@statkingclinical.com

Location: DocuSign

Signer Events

Baltazar Gomez-Mancilla

baltazar.gomez-mancilla@stalicla.com Security Level: Email, Account Authentication

(Required)

Signature

Maleul

Timestamp

Sent: February 18, 2022 | 08:57 Viewed: February 18, 2022 | 08:58 Signed: February 18, 2022 | 08:59

Signature Adoption: Drawn on Device

Signature ID:

78E6C319-C8F3-4E95-8414-A33B6E063709

Using IP Address: 92.140.206.228

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: August 13, 2021 | 11:17 ID: beebb2ce-daad-4f49-87c9-6b26dabb366a

Brian Kovacic

Brian@statkingclinical.com

Security Level: Email, Account Authentication

(Required)

Brian kovacic

Sent: February 18, 2022 | 08:57 Viewed: February 18, 2022 | 09:04 Signed: February 18, 2022 | 09:05

Signature Adoption: Pre-selected Style

Signature ID:

0E0504FA-2F53-4C14-AB39-2254119CC092 Using IP Address: 216.196.246.214

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):
I am the author of this document

Electronic Record and Signature Disclosure:

Accepted: February 18, 2022 | 09:04 ID: aed79dbf-95a8-4734-b136-5a5fa848032d

| Signer Events | Signature | Timestamp |
|---|---|---|
| Lori Christman | | Sent: February 18, 2022 08:57 |
| lori@statkingclinical.com | Lori Christman | Resent: February 18, 2022 10:08 |
| Senior Vice President | | Viewed: February 18, 2022 10:08 |
| Security Level: Email, Account Authentication (Required) | Signature Adoption: Pre-selected Style Signature ID: D32195A3-119A-4616-B959-EFE41655886B Using IP Address: 74.219.206.115 | Signed: February 18, 2022 10:09 |
| | With Signing Authentication via DocuSign password With Signing Reasons (on each tab): | |
| | I approve this document | |
| Electronic Record and Signature Disclosure:<br>Accepted: February 18, 2022 10:08<br>ID: 4adae6cc-21f4-4b6a-9455-3cc8b9262a35 | | |
| Mark Tetrick | 0 | Sent: February 18, 2022 08:57 |
| mtetrick@statkingclinical.com | male d. Tetrek | Viewed: February 18, 2022 08:57 |
| Clinical Trial Manager | | Signed: February 18, 2022 08:58 |

Signature Adoption: Uploaded Signature Image

FF75403B-BD93-466E-ABA9-DFBDFE59F935

With Signing Authentication via DocuSign password

Using IP Address: 216.196.246.214

Signature ID:

With Signing Reasons (on each tab):
I approve this document
Electronic Record and Signature Disclosure:

Statking Consulting, Inc.

(Required)

Security Level: Email, Account Authentication

Not Offered via DocuSign In Person Signer Events **Signature Timestamp Editor Delivery Events Status Timestamp Agent Delivery Events Status Timestamp Intermediary Delivery Events Status Timestamp Certified Delivery Events Status Timestamp Carbon Copy Events Status Timestamp** Witness Events **Signature Timestamp Notary Events Signature Timestamp Envelope Summary Events Status Timestamps** Hashed/Encrypted February 18, 2022 | 08:57 Envelope Sent Security Checked February 18, 2022 | 08:57 Certified Delivered Signing Complete Security Checked February 18, 2022 | 08:58 Completed Security Checked February 18, 2022 | 10:09 **Payment Events Status Timestamps Electronic Record and Signature Disclosure** 

# ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Statking Consulting, Inc. (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

# Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

# Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

# Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

# How to contact Statking Consulting, Inc.:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: mtetrick@statkingclinical.com

# To advise Statking Consulting, Inc. of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at mtetrick@statkingclinical.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

# To request paper copies from Statking Consulting, Inc.

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to mtetrick@statkingclinical.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with Statking Consulting, Inc.

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to mtetrick@statkingclinical.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

# Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

# Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send
  this Electronic Record and Disclosure to a location where you can print it, for future
  reference and access; and
- Until or unless you notify Statking Consulting, Inc. as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by Statking Consulting, Inc. during the course of your relationship with Statking Consulting, Inc..